## 来瑞特韦片治疗轻中型或重型新型冠状病毒感染 住院患者有效性的临床研究

# 病例报告表

| 版本号: | V 1.1 |
|------------|------------|
| 版本日期: | 2023年5月31日 |
| 中心名称: | |
| 中心号: | |
| 药物编号 | _ _ |
| 筛选号: | _ _ |
| 受试者姓名拼音缩写: | |

研究申办者:广州医科大学附属第一医院

#### 研究流程图

| 阶段 | 筛选期 | | | | | 治疗 | '期 | | | | | 随访 | i期 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 时间(天) | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 14 | 28 |
| 窗口期 | -2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | ±2 | ±4 |
| 知情同意书 | X | | | | | | | | | | | | |
| 入组/排除标准 | X | | | | | | | | | | | | |
| 人口统计学 1 | X | | | | | | | | | | | | |
| 个人史和过敏史 <sup>2</sup> | X | | | | | | | | | | | | |
| 病毒抗原检测3 | X | | | | | | | | | | | | |
| 新冠疫苗接种情况4 | X | | | | | | | | | | | | |
| 新冠病毒核酸检测5 | X | X | X | X | X | X | X | X | X | X | X | X* | X* |
| 胸部影像学检查6 | X | | | | | X* | | | | | X* | | X* |
| 血氧饱和度 7 | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 生命体征8 | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 临床症状 9 | X | X | X | Х | X | X | X | X | X | X | X | X | X |
| 体格检查 10 | X | X | X | Х | X | X | X | X | X | X | X | X | X |
| 实验室检查 11 | X | | | | | Х | | | | | X# | X# | |
| 炎性标志物 12 | X | | | | | X | | | | | X# | X# | |
| 治疗方案 13 | X | X | X | Х | X | Х | X | X | X | X | X | X | X |
| 合并用药 14 | X | X | X | Х | X | Х | X | Х | X | X | X | X | X |
| 安全性事件 15 | X | X | X | Х | X | Х | X | X | X | X | X | X | X |
| 疾病诊断信息 16 | X | X | X | Х | X | Х | X | X | X | X | X | X | X |
| 新冠病毒基因检测 17 | X | | | | | X | | | | | X | | |

注:

- a.\*为非必须,根据受试者身体情况,临床医生可酌情决定是否进行; #为出院前检查记录。
- b. 流感病毒检测、胸部影像学检查、实验室检查、炎症标记物等,签署知情前 5 天内的结果可以接受;检查报告如有异常临床意义(由研究医生判断),需在签署知情同意后,对异常项进行检测。
- c. 本研究拟定最长治疗期为 10 天,实际治疗期已受试者实际服药时间为准,受试者治疗期间(即转阴前)应每

日进行核酸检测并由研究者记录收集数据;若受试者转阴前即出院也将尽力收集受试者核酸检测结果至转阴,如却无办法收集也需要保证用药后 D10 的核酸检测及收集(如果受试者 D10 前仍未转阴);随访期即 D14 及 D28 核酸检测是否进行由研究者根据受试者回访时的症状进行相关判断,按需进行。

- 1) 人口统计学包括:年龄、性别、民族、出生日期等;
- 2) 个人史和过敏史包括:既往病史、既往新冠病史、吸烟饮酒情况及药物过敏史等;
- 3) 病毒抗原检测包括:甲型/乙型流感病毒抗原或核酸检测;
- 4) 新冠疫苗接种情况包括:疫苗种类、接种时间、次剂、厂家等;
- 5) 新冠病毒核酸检测包括:标本类型、结果、Ct 值、ORF1ab 基因 Ct 值、N 基因 Ct 值、抗原检测结果等;(优选每天进行核酸检测)
- 6) 胸部影像学检查包括胸部 CT 或胸片;
- 7) 血氧饱和度:指脉氧饱和度;
- 8) 生命体征;体温、呼吸、血压、脉搏等;
- 9) 新型冠状病毒感染相关临床症状:包括鼻塞或流涕、咽痛、呼吸短促或呼吸困难、咳嗽、乏力、肌肉或身体疼痛、头痛、寒战、发热、恶心、呕吐、腹泻、嗅觉减退、味觉减退等;
- 10) 体格检查:一般状况、头颈部、胸部、腹部、脊柱和四肢关节、神经系统、皮肤、淋巴、精神状态等;
- 11) 实验室检查包含血常规、血生化、凝血功能、动脉血气、血脂;
- a. 血常规: 红细胞计数、血红蛋白、血小板计数、白细胞计数、红细胞压积、中性粒细胞计数和淋巴细胞计数;
- b. 血生化: 丙氨酸氨基转移酶、门冬氨酸氨基转移酶、碱性磷酸酶、总胆红素、直接胆红素、总蛋白、白蛋白、 尿素氮、肌酐、血糖、尿酸等;
- c. 凝血功能: 凝血酶原时间、活化部分凝血活酶时间、纤维蛋白原、凝血酶时间、D-二聚体。
- d. 动脉血气分析: 氧饱和度、二氧化碳分压、氧分压、碳酸氢、氧合指数;
- e. 血脂: 总胆固醇、甘油三酯、高密度脂蛋白、低密度脂蛋白;
- 12) 炎症标志物: C 反应蛋白、降钙素原;
- 13) 治疗方案:包括研究期间治疗新冠用药及相关非用药干预方式记录(吸氧、机械通气等);
- 14) 合并用药:治疗过程中产生的"治疗方案"部分未记录的药物应用详情;
- 15) 安全性事件:记录不良事件及严重不良事件;
- 16) 疾病诊断信息:确诊方式、临床分型、脓毒症诊断、是否住院、ICU、死亡等。
- 17)新冠病毒基因检测:基线病毒分型及耐药突变分析,如在第5天、第10天病毒核酸已转阴,则使用最后一次病毒可测时间点的标本。

#### 在正式填表前,请认真阅读以下说明

#### 病例收集表填表说明

- 1. 病例收集表的每一页都须完成,所有的项目均应填写。选用钢笔或签字笔用力填写表格。在"□"处填入"√"或"×"表示选择此项,例: ☑/区。如果此项"未做"则填入"ND"; "不详"则填入"NK"; "不适用"则填入"NA",所有选择等级的数字,填入"□"内,例: □4□。
- 2. 填写务必认真、准确、清晰、如实,不能随意涂改,如填写确有错误,修改时不能涂 黑或使用涂改液,应将填写错误的数据用横线居中划出,在旁边写上正确的数据,并 由负责医师在修改处签名、注明日期。例如: 24 28 套覆 2002-12-12
- 3. 患者姓名拼音缩写需填满四格,两字姓名分填两字前两个字母,三字姓名填前两字首字母与第三字前两个字母,四字姓名填每字首字母。举例:

| 张红 | Z | Н | Н | 0 | 李淑明 | L | S | M | Ι | 欧阳小惠 | 0 | Y | X | Н |
|----|---|---|---|---|-----|---|---|---|---|------|---|---|---|---|
|----|---|---|---|---|-----|---|---|---|---|------|---|---|---|---|

严格观察和如实填写不良反应记录表。记录不良反应的发生时间、严重程度、持续时间、采取的措施和转归。

### 访视1-筛选期(入组前2天)

| 入组/排除标准 |
|-----------------------------------------------------|
| │<br>│□研究前签署知情同意书、并对研究内容、过程及可能出现的不良反应充分了解; |
| <br> □年龄≥18岁,性别不限; |
| │<br>│□症状:至少有以下 14 项症状中的 1 项:鼻塞或流涕、咽痛、呼吸短促或呼吸困难、咳嗽 |
| 乏力、肌肉或身体疼痛、头痛、寒战、发热、恶心、呕吐、腹泻、嗅觉减退、味觉减退。 |
| □入组前 120h 内经鼻咽拭子检测确诊新型冠状病毒感染,新型冠状病毒核酸检测 Ct 值≤3 |
| (QPCR, ORF1ab 基因或 N 基因的 Ct 值≤30); |
| □符合以下疾病分型和病程(符合 A、B、C 中任意一条即可): |
| ► A. 轻、中型新型冠状病毒感染的住院患者且不伴有任一高危风险因素; 危风险因素有 |
| 年龄≥65岁;未接种新冠疫苗;患有慢性疾病(心血管疾病、肾病、呼吸系统疾病、 |
| 糖尿病、神经认知障碍等);各种形式的免疫抑制剂人群(肿瘤放化疗、器官或造血干 |
| 细胞移植、先天性免疫缺陷、HIV 感染、激素/免疫抑制剂/生物制剂使用者等);肥原 |
| (BMI≥30); |
| ▶ B. 轻、中型新型冠状病毒感染伴有任一高危风险因素的住院患者,且发病(出现 14 耳 |
| 症状中至少一项)5天(不含)以上;高危风险因素同A。 |
| ➤ C. 重型新型冠状感染住院患者。符合下列任何一条: 1)呼吸窘迫, RR≥30 次/分; 2) 青 |
| 息状态下,指氧饱和度≤93%;3)动脉血氧分压(PaO2)/吸氧浓度(FiO2)≤300mmHg; 临 |
| 床症状进行性加重,肺部影像学显示 24~48 小时内病灶明显进展>50%者; |
| □同意在整个研究期间至停药后3个月内采取有效避孕措施。 |
| 排除标准(受试者不能满足以下任一排除标准): |
| │<br>│□对来瑞特韦片成分或任何辅料过敏患者 <b>;</b> |

□发病 5 天内伴任一高危风险因素人群轻、中型新冠感染的住院患者(高危风险因素同纳入

| A); |
|------------------------------------------------|
| □危重型新型冠状病毒感染患者;。危重型患者为符合以下情况之一者:出现呼吸衰竭,且 |
| 需要机械通气; 出现休克; 合并其他器官功能衰竭需 ICU 监护治疗; |
| □重度肾损伤患者(Ccr <30 mL/min); |
| □患有精神疾患的患者; |
| □昏迷、吞咽困难患者; |
| □筛选时明显的肝功异常(ALT 或 AST≥10 ULN,或总胆红素≥2 ULN); |
| □HIV-1 感染未得到控制的患者; |
| □甲型/乙型流感病毒抗原或核酸阳性的患者; |
| □入组前 28 天内及计划在研究期间接种疫苗者; |
| □妊娠、哺乳期女性或妊娠试验阳性者; |
| □在用药前 1 个月内参加并接受其他临床试验药物者; |
| □依从性差,不能配合完成试验; |
| □本次病程中使用过或在研究期间计划使用过抗新型冠状病毒药物(如 Paxlovid、阿兹夫定、 |
| 安巴韦单抗/罗米司韦单抗注射液、静注 COVID-19 人免疫球蛋白或新冠康复者恢复期血浆 |
| 等); |
| □医生认为其它不适合入组的情况。 |
| 一、人口统计学 |
| 出生日期: _ - _ - _ (yyyy-mm-dd) |
| 年龄: 岁 |
| 性别: □男 □女 |
| 民族:□汉族 □其他,请说明: |
| 婚姻状况:□未婚 □已婚 □离异 □丧偶 |
| 教育程度:□小学及以下 □初中及以下 □高中及以下 □大学及以上 |
| 职业类型:□无业 □学生 □脑力劳动者 □体力劳动者 □其他 |
| 二、个人史和过敏史 |
| 是否有疾病史:□是 □否 |

| 如"是"),疾病种类:□心脏病 □慢性肺病 □糖尿病 □血红蛋白病 | □免疫抑 |
|---|---|
| 状态 □透析 □肝病 □肾病 □代谢性疾病 □神经系疾病 □肿瘤 | |
| 其他疾病史 | |
| 是否有新型冠状病毒感染史:□是 □否 | |
| (如"是"),是否住院:□是□□否 | |
| 吸烟史:□从未吸烟 □目前吸烟 □已戒烟 | |
| (如"目前吸烟"),每天吸烟数量:支 | |
| 饮酒史:□从未饮酒 □目前饮酒 □已戒酒 | |
| (如"目前饮酒"),饮酒频率:□每周1次 □每周2-3次 □每周4-5次 | □几乎每 |
| 天 | |
| 是否有药物滥用史:□是 □否 | |
| 是否有药物过敏史: □是 □否 | |
| (如"是")药物名称:; 反应类型/表现: | |
| 三、病毒抗原检测 | |
| 注: 抗原或核酸检测均可,进行哪一项则勾选哪一项 | |
| │<br>│ 是否进行甲型/乙型流感病毒抗原检测: □是 □否 | |
| 如"否"请勾选未做项:□甲流 □乙流 | |
| 如 "否"请勾选未做项: □甲流 □乙流<br> 检测日期: _ - - (yyyy-mm-dd) | |
| 检测日期: _ _ - - (yyyy-mm-dd) | |
| 检测日期: _ - - (yyyy-mm-dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 | |
| 检测日期: _ _ - - (yyyy-mm-dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 乙型流感病毒抗原检测结果: □阴性 □阳性 | |
| 检测日期: _ _ - - (yyyy-mm-dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 乙型流感病毒抗原检测结果: □阴性 □阳性 是否进行甲型/乙型流感病毒核酸检测: □是 □否 | |
| 检测日期: _ _ - - - (yyyy¬mm¬dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 乙型流感病毒抗原检测结果: □阴性 □阳性 是否进行甲型/乙型流感病毒核酸检测: □是 □否 如"否"请勾选未做项: □甲流 □乙流 | |
| 检测日期: _ _ - - _ (yyyy-mm-dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 乙型流感病毒抗原检测结果: □阴性 □阳性 是否进行甲型/乙型流感病毒核酸检测: □是 □否 如"否"请勾选未做项: □甲流 □乙流 检测日期: _ _ - - (yyyy-mm-dd) | |
| 检测日期: _ _ - - _ - _ (yyyy-mm-dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 乙型流感病毒抗原检测结果: □阴性 □阳性 是否进行甲型/乙型流感病毒核酸检测: □是 □否 如"否"请勾选未做项: □甲流 □乙流 检测日期: _ - _ - _ - _(yyyy-mm-dd) 甲型流感病毒核酸检测结果: □阴性 □阳性 | |
| 检测日期: _ - - - (yyyy-mm-dd) 甲型流感病毒抗原检测结果: □阴性 □阳性 乙型流感病毒抗原检测结果: □阴性 □阳性 是否进行甲型/乙型流感病毒核酸检测: □是 □否 如 "否"请勾选未做项: □甲流 □乙流 检测日期: _ - - (yyyy-mm-dd) 甲型流感病毒核酸检测结果: □阴性 □阳性 乙型流感病毒核酸检测结果: □阴性 □阳性 | |

| □未接种 | | | | |
|------------------------|---------------|----------|--------|-------|
| □第一针,时间 _ _ - _ - _ | _ - (yy | yy-mm-do | d) | |
| 疫苗厂家:□北京生物 □北京科兴 | □武汉生物 □ | 康希诺 | □智飞龙科马 | □长春祁健 |
| □其他 | | | | |
| □第二针,时间 _ _ - - | _ - (yyy | y-mm-dd) | ) | |
| 疫苗厂家:□北京生物 □北京科兴 | □武汉生物 □ | 康希诺 | □智飞龙科马 | □长春祁健 |
| □其他 | | | | |
| □第三针,时间 _ _ - - | _ - (yyy | y-mm-dd) | ) | |
| 疫苗厂家:□北京生物 □北京科兴 | □武汉生物 □ | 康希诺 | □智飞龙科马 | □长春祁健 |
| □其他 | | | | |
| □第四针,时间 _ _ - _ - _ | _ - (yy | yy-mm-do | d) | |
| 疫苗厂家:□北京生物 □北京科兴 | □武汉生物 □ | 康希诺 | □智飞龙科马 | □长春祁健 |
| □其他 | | | | |
| 五、亲 | <b>听冠病毒核酸</b> | 趁检测 | | |
| 是否进行新冠病毒核酸检测:□是 □ | ]否 | | | |
| 检测日期: _ _ - _ - _ - | _ (yyyy-m | m-dd) | | |
| 标本类型:□鼻咽拭子□□咽拭子 | | | | |
| 采样日期: _ _ - - | _ (yyyy-m | m-dd) | | |
| 新型冠状病毒 ORF1ab 基因: □阴性 | □阳性 | | | |
| 新型冠状病毒 ORF1ab 基因 Ct 值: | | | | |
| 新型冠状病毒 N 基因: □阴性 □阳 | 性 | | | |
| 新型冠状病毒 N 基因 Ct 值: | | | | |
| 六、 | 胸部影像学 | 检测 | | |
| 是否进行胸部影像检查:□是□□否 | | | | |
| 检查日期: _ _ - - | _ (yyyy-m | m-dd) | | |
| 检查名称 | 检查内容 | | 临床意义 | |
| 協立! / | | 口正 | 常 □昇常ラ | E临床意义 |
| 胸部(肺部)CT | | □异 | 常有临床意义 | □未查 |

| Ba da / 日本 da / y 自 | 444 | | □正常 □异常无临床意义 |
|---|---|---|---|
| 胸部(肺部)X身 | 引线 | | □异常有临床意义 □未查 |
| | 七、 | 血氧饱和 | 度 |
| 是否进行血氧饱和度检查 | <b>:</b> □是 □否 | | |
| 检查日期: _ _ | . - - | (yyyy-n | nm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| <b>化</b> | | % | □正常 □异常无临床意义 |
| 指端脉氧饱和度 | | % | □异常有临床意义 □未查 |
| | 八、 | 生命体征 | E |
| 是否进行生命体征检查: | □是 □否 | | |
| 检查日期: _ _ | - - | (yyyy-n | nm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 体温 | | $^{\circ}$ | □正常 □异常无临床意义 |
| , , am. | | | □异常有临床意义 □未查 |
| <br> 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 呼吸频率 | | 次/分 | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 血压 (收缩压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| | 九、 | 临床症状 | <del>\text{\tin}\text{\tett{\text{\tetx{\text{\ti}\tint{\text{\text{\text{\tin}\tint{\text{\text{\text{\text{\ti}\tint{\text{\text{\texi}\tinz{\text{\texit{\texi}\tinz{\text{\texi}\text{\text{\texit{\texit{\texit{\texi}\tint{\texit{\texi{\ti}\tint{\texit{\texi{\texi{\texi{\texi}\texit{\texi{\texi{</del> |
| 是否有新冠感染相关临床 | 症状:□是 | □否 | |
| (如"是"),临床症状:[ | □鼻塞或流涕 | □咽痛 □ | ]呼吸短促或呼吸困难 □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | ]寒战 [ | ]发热 □恶心 □呕吐 □腹泻 |
| □嗅觉减退□呀 | 总觉 减 退 | □其他症 | 【状:开始日期: |
| _ _ - - | - (yyyy- | mm-dd) | |
| 结束日期: | | | |

| 十、体格检查 | | | | |
|---|---|---|---|---|
| 是否进行体格检查:□是 | □否 | | | |
| 检查日期: | - - _ | (yyyy-r | nm-dd) | |
| 检查项目 | ı | 临床意义 | | 若有异常,请描述 |
| 一般情况 | □正常 □ | | | |
| 头颈部 | □正常 □ | | | |
| 胸部 | □正常 □ | | | |
| 腹部 | □正常 □ | | | |
| 脊柱和四肢关节 | □正常 □ □ □ 异常有临床 | | | |
| 神经系统 | □正常 □ □ □ 异常有临床; | | | |
| 皮肤 | □正常 □ | | | |
| 淋巴 | □正常 □ | | 意义<br>未查 | |
| 其他 | □正常 □ | | | |
| | +-, | 实验室检 | <b>全</b> | |
| 是否进行血常规检查:□ | 是□否 | | | |
| 检查日期: _ - - - | _ _ - (yyy | y-mm-dd) | | |
| 检查项目 | 检查结果 | 单位 | | 临床意义 |
| 红细胞计数(RBC) | | 10 <sup>12</sup> /L | □正常<br>□异常有临 | □异常无临床意义<br>5床意义 □未查 |

| 自细胞计数(WBC) | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
|---|---|---|---|
| 白细胞的数(WBC) | | 10 /L | □异常有临床意义 □未查 |
| 血红蛋白(Hb) | | g/L | □正常 □异常无临床意义 |
| 皿红斑口(110) | | g/L | □异常有临床意义 □未查 |
| 血小板计数(PLT) | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
| 皿刀切以 致 (111) | | 10 /L | □异常有临床意义 □未查 |
| <br> | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
| 717日土7里5山月201 安久 | | 10 /L | □异常有临床意义 □未查 |
| <br> 红细胞压积(HCT)) | | % | □正常 □异常无临床意义 |
| 红细胞压然(nci)) | | 70 | □异常有临床意义 □未查 |
| 淋巴细胞计数(Lym) | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
| | | 10 <sup>7</sup> /L | □异常有临床意义 □未查 |
| 是否进行血生化检查:□ | 是□否 | | |
| 检查日期: _ _ _ - - - | _ _ - (yyy | y-mm-dd) | |
| 检查项目 | 检查结果 | 単位 | 临床意义 |
| | 检查结果<br>———————————————————————————————————— | 単位<br>□U/L | 临床意义<br>□正常 □异常无临床意义 |
| 检查项目<br>谷丙转氨酶(ALT) | 检查结果<br> | | |
| 谷丙转氨酶(ALT) | 检查结果 | □U/L | □正常 □异常无临床意义 |
| | 检查结果 | □U/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 谷丙转氨酶(ALT)<br>谷草转氨酶(AST) | 检查结果 | □U/L □IU/L □U/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 |
| 谷丙转氨酶(ALT) | 检查结果 | □U/L □IU/L □U/L □IU/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 □未查 □异常无临床意义 □未查 |
| 谷页转氨酶(ALT) 谷草转氨酶(AST) 碱性磷酸酶(ALP) | 检查结果 | □U/L □IU/L □IU/L □U/L □U/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 □未查 □异常无临床意义 □未查 □异常有临床意义 □未查 □正常 □异常无临床意义 |
| 谷丙转氨酶(ALT)<br>谷草转氨酶(AST) | 检查结果 | □U/L □IU/L □IU/L □U/L □IU/L □IU/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 □未查 □异常无临床意义 □未查 □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 谷丙转氨酶(ALT) 谷草转氨酶(AST) 碱性磷酸酶(ALP) | 检查结果 | □U/L □IU/L □IU/L □U/L □IU/L □IU/L □umol/L | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 谷页转氨酶(ALT) 谷草转氨酶(AST) 碱性磷酸酶(ALP) | 检查结果 | □U/L □IU/L □IU/L □U/L □IU/L □IU/L □umol/L □mg/dl | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 谷丙转氨酶(ALT) 谷草转氨酶(AST) 碱性磷酸酶(ALP) | 检查结果 | □U/L □IU/L □IU/L □IU/L □IU/L □IU/L □umol/L □umol/L □umol/L | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |

| 白蛋白(ALB) | | α/Ι | □正常 □异常无临床意义 |
|---|---|---|---|
| 口虫口(ALD) | | g/L | □异常有临床意义 □未查 |
| 尿素氮(BUN) | | o 1/I | □正常 □异常无临床意义 |
| / | | mmol/L | □异常有临床意义 □未查 |
| 血肌酐 (Cr) | | □mg/dl | □正常 □异常无临床意义 |
| (急性肾衰 □是□否) | | □umol/L | □异常有临床意义 □未查 |
| de la | | 1/7 | □正常 □异常无临床意义 |
| 血糖(Glu) | | mmol/L | □异常有临床意义 □未查 |
| | | 1.77 | □正常 □异常无临床意义 |
| 尿酸(UA) | | μmol/L | □异常有临床意义 □未查 |
| <u>Е</u> Ш (Т/) | | 1/T | □正常 □异常无临床意义 |
| 钾 (K) | | mmol/L | □异常有临床意义 □未查 |
| Eth(NI <sub>2</sub> ) | | | □正常 □异常无临床意义 |
| 钠(Na) | | mmol/L | □异常有临床意义 □未查 |
| 氯(Cl) | | mmol/L | □正常 □异常无临床意义 |
| ऋ( (СГ) | | IIIIIIOI/L | □异常有临床意义 □未查 |
| 是否进行凝血功能检查: | □是 □否 | | |
| 检查日期: - | _ _ - (yyy | yy-mm-dd) | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 海南南百叶河(PT) | | _ | □正常 □异常无临床意义 |
| 凝血酶原时间(PT) | | S | □异常有临床意义 □未查 |
| 活化部分凝血活酶时间 | | | □正常 □异常无临床意义 |
| (APTT) | | S | □异常有临床意义 □未查 |
| 纤维蛋白原(Fg) | | □g/L | □正常 □异常无临床意义 |
| 月採虫口凉(Fg) | | □mg/dl | □异常有临床意义 □未查 |
| 凝血酶时间(TT) | | G | □正常 □异常无临床意义 |
| 7次、川山日本日1月日(111) | | S | □异常有临床意义 □未查 |
| D-二聚体(D-Dimer) | | □ µ g/L | □正常 □异常无临床意义 |

| | | □mg/L | □异常有临床意义 □未查 |
|---|---|---|---|
| 是否进行动脉血气分析检 | 测:□是 □ | 否 | , |
| 检查日期: _ _ - - | _ _ - (yyy | y-mm-dd) | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| *** | | | □正常 □异常无临床意义 |
| pН | | | □异常有临床意义 □未查 |
| 电复数和度 | | 0/ | □正常 □异常无临床意义 |
| 血氧饱和度 | | % | □异常有临床意义 □未查 |
| 一复从理八耳(P-CO) | | | □正常 □异常无临床意义 |
| 二氧化碳分压(PaCO <sub>2</sub> ) | | mmHg | □异常有临床意义 □未查 |
| 复八厂 ( <b>P-O</b> ) | | | □正常 □异常无临床意义 |
| 氧分压(PaO <sub>2</sub> ) | | mmHg | □异常有临床意义 □未查 |
| 型形气(HCO-) | | /T | □正常 □异常无临床意义 |
| 碳酸氢(HCO <sub>3</sub> -) | | mg/L | □异常有临床意义 □未查 |
| 氧合指数(PaO <sub>2</sub> /FiO <sub>2</sub> ) | | mmHa | □正常 □异常无临床意义 |
| 車(□1目刻(PaO2/FIO2) | | mmHg | □异常有临床意义 □未查 |
| 是否进行血脂检测:□是 | □否 | | |
| 是否进行血脂检测:□是<br>检查日期:□□□□□-□ | | y-mm-dd) | |
| | | y-mm-dd)<br>单位 | 临床意义 |
| 检查日期: _ - -<br>检查项目 | _ _ - _ (yyy | | 临床意义<br>□正常 □异常无临床意义 |
| 检查日期: _ - - | _ _ - _ (yyy | 单位 | |
| 检查日期: _ - -<br>检查项目<br>总胆固醇(TC) | _ _ - _ (yyy | 单位 | □正常 □异常无临床意义 |
| 检查日期: _ - -<br>检查项目 | _ _ - _ (yyy | 单位<br>mmol/L | □正常 □异常无临床意义 □未查 |
| 检查日期: _ - - - - | _ _ - _ (yyy | 单位<br>mmol/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 |
| 检查日期: _ - -<br>检查项目<br>总胆固醇(TC) | _ _ - _ (yyy | 单位<br>mmol/L<br>mmol/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 □未查 □异常无临床意义 □未查 |
| 检查日期: _ - - - | _ _ - _ (yyy | 单位<br>mmol/L<br>mmol/L | □正常 □异常无临床意义 □未查 □正常 □异常无临床意义 □未查 □异常无临床意义 □未查 □异常有临床意义 □未查 □正常 □异常无临床意义 |
| 检查日期: _ - - - - | _ _ - _ (yyy | 单位<br>mmol/L<br>mmol/L | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 检查日期: _ - - - | _ - (yyy<br>检查结果 | 单位<br>mmol/L<br>mmol/L | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 检查日期: _ - - - - - - - | _ - (yyy<br>检查结果<br>是 □否 | 单位<br>mmol/L<br>mmol/L | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 检查日期: _ - | _ - (yyy<br>检查结果<br>是 □否 | 单位<br>mmol/L<br>mmol/L<br>mmol/L | □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 |

| | | □IU/ml | □异常有临床意义 □未查 |
|---|---|---|---|
| 无旺於休 (HOV) | | □S/CO | □正常 □异常无临床意义 |
| 丙肝抗体(HCV) | | □IU/ml | □异常有临床意义 □未查 |
| 梅毒体 | | S/CO | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查<br>□正常 □异常无临床意义 |
| HIV 抗体 | | S/CO | □□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ |
| | 十二、 | 炎症标志 | ·<br>法物 |
| 是否进行炎症标志物检查 | <b>:</b> □是 □否 | ; | |
| 检查日期: _ - - - | _ _ - (yyy | yy-mm-dd) | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| | | □ µ g/L | |
| C 反应蛋白 | | □mg/dl | □正常 □异常无临床意义 |
| | | □mg/L | - □异常有临床意义 □未查 |
| | | | □正常 □异常无临床意义 |
| 降钙素原 | 降钙素原 ng/ml | | □异常有临床意义 □未查 |
| | 十三 | 、治疗方 | 案 |
| 新冠感染药物治疗 | | | |
| 来瑞特韦给药情况 | | | |
| 药物规格: mg | | | |
| 初始给药日期: _ - - (yyyy-mm-dd) | | | |
| 是否持续:□是 □否 | | | |
| 结束给药日期: _ _ - - (yyyy-mm-dd) | | | |
| 给药剂量: mg | | | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | | | |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | | | |
| 注射 □其他 | | | |
| 总剂量: mg | | | |

| 其他新冠治疗药物给药情况 |
|-------------------------------------------------|
| 抗病毒小分子药物 |
| 药物名称:□奈玛特韦片/利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 初始给药日期: _ - - (yyyy-mm-dd)<br>是否持续: □是 □否 |
| <br> 是否持续: □是 □否 |
| 是否持续: □是 □否 □ |
| 是否持续: □是 □否 |
| 是否持续: □是 □否 |
| 是否持续: □是 □否 |
| 是否持续: □是 □否 |
| 是否持续: □是 □否 |
| 是否持续: □是 □否 |

| 是否持续:□是 □否 |
|-------------------------------------------------|
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |

| 如"是"请勾选:□有创 □无创 |
|------------------------------------------------------------|
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 十四、合并用药 |
| 是否发生合并用药:□是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 |
| □抗生素:□抗真菌类 □抗病毒类 |
| □糖皮质激素 |
| 日期: _ _ - - - (yyyy-mm-dd) 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 十五、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: _ _ - - (yyyy-mm-dd) |
| 注:如有不良事件,请记录在"不良事件记录表" |
| 十六、疾病诊断信息 |
| 是否确诊新型冠状病毒感染:□是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| <br> 是否出院: □是 □ □否 |

| 出院日期: _ - - (yyyy-mm-dd) |
|---------------------------------|
| 是否死亡: □是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |
| 十七、新冠病毒基因检测 |
| 是否保留受试者新冠病毒核酸检测样本:□是□□否 |
| 标本类型:□鼻拭子 □咽拭子 |

## 访视 2-治疗期 (第1天)

| 访视日期: | <u> </u> | - | - | <b>(</b> y) | /yy-mm-dd) |
|-------|----------|---|---|-------------|------------|
|-------|----------|---|---|-------------|------------|

| 一、新冠病毒核酸检测 | | | |
|---|---|---|---|
| 是否进行新冠病毒核酸检测:□是□□否 | | | |
| 检测日期: _ | _ - _ - | (yyyy-m | m-dd) |
| 标本类型:□鼻咽扭 | 式子 □□咽拭子 | | |
| 采样日期: | _ - _ | (yyyy-m | mm-dd) |
| 新型冠状病毒 ORF1a | ab 基因: □阴性 □ | 阳性 | |
| 新型冠状病毒 ORF1a | ab 基因 Ct 值: | _ | |
| 新型冠状病毒N基因 | 因:□阴性 □阳性 | | |
| 新型冠状病毒N基因 | 因 Ct 值: | | |
| | =, ] | 血氧饱和 | 度 |
| 是否进行血氧饱和原 | 度检查:□是□□否 | | |
| 检查日期: | _ - _ | (yyyy-m | mm-dd) |
| 检查项目 | 检查结果 単位 临床意义 | | 临床意义 |
| 指端脉氧饱和度 | | % | □正常 □异常无临床意义 |
| 1日师/// 刊(巴作/文 | | 70 | □异常有临床意义 □未查 |
| 三、生命体征 | | | |
| 是否进行生命体征检查:□是 □否 | | | |
| 检查日期: _ - _ - _ (yyyy-mm-dd) | | | |
| 检查项目 检查结果 单位 临床意义 | | | |
| 体温 | | °C | □正常 □异常无临床意义 |
| 77 m. | | | □异常有临床意义 □未查 |
| 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 呼吸频率 次/分 □正常 □异常无临床意义 | | | |

| | | | □异常有临床意义 □未查 |
|---|---|---|---|
| 血压(收缩压) | | mmHg | □正常 □异常无临床意义 |
| 皿压(収細压) | | IIIIIII | □异常有临床意义 □未查 |
| 血压(舒张压) | | mmHg | □正常 □异常无临床意义 |
| III.ZE (B) JKZE/ | | 111111111111111111111111111111111111111 | □异常有临床意义 □未查 |
| | 四、 | 临床症状 | 比 |
| 是否有新冠感染相关临床 | 症状:□是 □ | ]否 | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | □呼吸短促或呼吸困难 □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 [ | □发热 □恶心 □呕吐 □腹泻 |
| □嗅觉减退 □味觉减过 | 艮 □其他症状 | : | |
| 开始日期: _ _ | - _ - _ | _ (уууу- | mm-dd) |
| 结束日期: _ _ | - - | _ (уууу- | -mm-dd) |
| | 五、 | 体格检查 | 查 |
| 是否进行体格检查:□是 □否 | | | |
| 检查日期: _ _ | - - | _ (уууу- | -mm-dd) |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常□! | 异常无临床 | E意义 |
| /X1770 | □异常有临床意 | :义 □ | 1未查 |
| <br> 头颈部 | □正常 □⅓ | 异常无临床 | 意义 |
| | □异常有临床意 | :义 🗆 | ]未查 |
| <br> 胸部 | □正常□⅓ | 异常无临床 | 意义 |
| 7,4,4,11 | □异常有临床意 | :义 □ | ]未查 |
| 腹部 | □正常 □⅓ | 异常无临床 | 意义 |
| 4η δη | □异常有临床意 | :义 □ | ]未查 |
| 脊柱和四肢关节 | □正常 □፶ | 异常无临床 | 意义 |
| 有任和四放大月 | □异常有临床意 | :义 □ | ]未查 |
| ÷中//2 ヹ レント | □正常 □⅓ | 异常无临床 | 意义 |
| 神经系统 | □异常有临床意 | :义 □ | ]未查 |
| 皮肤 | □正常 □臭 | 异常无临床 | 意义 |

| | □异常有临床意义 □未查 |
|---|---|
| 淋巴 | □正常 □异常无临床意义 |
| | □异常有临床意义 □未查 |
| 11.71 | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| <br> 药物规格: _ mg | |
| 初始给药日期: _ | 初始给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否持续: □是 □否 | |
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) | |
| 给药剂量: mg | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情况 | |
| 抗病毒小分子药物 | |
| 药物名称: □奈玛特韦片/利托那韦片 (Paxlovid) □先诺特韦片/利托那韦片 (先诺欣) | |
| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 | |
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ - _ - _ - (yyyy-mm-dd) | |
| 是否持续: □是 □否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| <br> 给药途径: □□服 □♬ | 引部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 □ |

| 注射 □其他 |
|-----------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称:□COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|---|
| 结束给药日期: _ - _ - _ - _ (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持:□是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药: □是 □否 |
| 如"是"请在此处做药物分类勾选: □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 □抗生素:□抗真菌类 □抗病毒类 □糖皮质激素 □期: _ _ - _ - _ (yyyy-mm-dd) |
| 注:如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 是否发生安全性事件: □是 □否 |
| 日期: |

| 注: 如有不良事件,请记录在"不良事件记录表" |
|----------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - _ (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

## 访视 3-治疗期 (第2天)

| 访视日期: <br> | - - - | _ (yyyy-r | mm-dd) |
|---------------------------------|---------------|------------|---------------|
| | 一、新冠 | 病毒核酢 | <b>发检测</b> |
| 是否进行新冠病毒核 | 亥酸检测:□是 □否 | | |
| 检测日期: _ | _ - - | _ (уууу- | mm-dd) |
| 标本类型:□鼻咽拮 | 战子 □□咽拭子 | | |
| 采样日期: _ | _ - - | _ (уууу- | mm-dd) |
| 新型冠状病毒 ORF1a | ab 基因: □阴性 □阝 | 阳性 | |
| 新型冠状病毒 ORF1a | ab 基因 Ct 值: | - | |
| 新型冠状病毒 N 基团 | 団:□阴性 □阳性 | | |
| │<br>│新型冠状病毒 N 基团 | 因 Ct 值: | | |
| | 二、1 | 血氧饱和 | 度 |
| 是否进行血氧饱和原 | 度检查:□是□□否 | | |
| 检查日期: - - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| <br> 指端脉氧饱和度 | | % | □正常 □异常无临床意义 |
| 1日2冊が主(地7円)支 | | | □异常有临床意义 □未查 |
| 三、生命体征 | | | |
| 是否进行生命体征核 | 佥查:□是□□否 | | |
| 检查日期: _ - - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 体温 | | °C | □正常 □异常无临床意义 |
| 17 1111 | | | □异常有临床意义 □未查 |
| <br> 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| )41 <b>-1</b> 74 | | | □异常有临床意义 □未查 |

次/分

呼吸频率

□正常

□异常无临床意义

| | | | □异常有临床意义 □未查 |
|---|---|---|---|
| | | | 71.11.14.11.11.11.11.11.11.11.11.11.11.11 |
| <br> 血压(收缩压) | mmHg | mmHg | □正常 □异常无临床意义 |
| | | □异常有临床意义 □未查 | |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 |
| III./II. (II.) (IV.II.) | | | □异常有临床意义 □未查 |
| | 四、 | 临床症状 | 犬 |
| 是否有新冠感染相关临床 | 症状:□是 [ | □否 | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | □呼吸短促或呼吸困难 □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 | □发热 □恶心 □呕吐 □腹泻 |
| │ □嗅觉减退 □味觉减退 | 艮 □其他症状 | : | |
| 开始日期: _ | - - | _ (уууу- | mm-dd) |
| 结束日期: | - - | _ (уууу- | mm-dd) |
| | 五、 | 体格检查 | 查 |
| 是否进行体格检查:□是 | □否 | | |
| 检查日期: | - - | _ (yyyy- | mm-dd) |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常□! | 异常无临床 | 意义 |
| AX IA VII | □异常有临床意 | 义 □ | 未查 |
| <br> 头颈部 | □正常 □! | 异常无临床 | 意义 |
| | □异常有临床意义 □未査 | | |
| 胸部 | □正常□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ | 异常无临床 | 意义 |
| 加加可 | □异常有临床意义 □未查 | | |
| 腹部 | □正常 □! | 异常无临床 | 意义 |
| 川文 口中 | □异常有临床意 | :义 □ | 未查 |
| 脊柱和四肢关节 | □正常 □! | 异常无临床 | 意义 |
| | □异常有临床意 | :义 □ | 未查 |
| 沖瓜 互 ひ | □正常□! | 异常无临床 | 意义 |
| 神经系统 | □异常有临床意 | :义 □ | 未查 |
| 皮肤 | □正常□! | 异常无临床 | 意义 |

| | □异常有临床意义 □未查 |
|---|---|
| 淋巴 | □正常 □异常无临床意义 |
| | □异常有临床意义 □未查 |
| | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: _ mg | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |
| 总剂量: _ mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氚瑞米德韦片(仁 | |
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ _ - - (yyyy-mm-dd) | |
| 是否持续: □是 □否 | |
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径:□□服 □周 | 局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |

| 注射 □其他 |
|-----------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称: □连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| <br> 初始给药日期: - - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|-------------------------------------------------|
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药: □是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 |
| □抗生素: □抗真菌类 □抗病毒类 □糖皮质激素 |
| 日期: _ _ - - (yyyy-mm-dd) |
| 注:如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: - - (yyyy-mm-dd) |

| 注: 如有不良事件,请记录在"不良事件记录表" |
|----------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - _ (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

#### 访视 4-治疗期 (第3天)

访视日期: |\_\_|\_|-|\_-|-|(yyyy-mm-dd) 一、新冠病毒核酸检测 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_\_|\_\_|-|\_\_|-|\_\_|-|(yyyy-mm-dd) 标本类型:□鼻咽拭子□□咽拭子 采样日期: |\_\_|\_|\_|-|\_\_|-|\_|-|(yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、血氧饱和度 是否进行血氧饱和度检查:□是□□否 检查日期: | | | | |-| | | (yyyy-mm-dd) 单位 检查项目 检查结果 临床意义 □正常 □异常无临床意义 指端脉氧饱和度 % □异常有临床意义 □未查 三、生命体征 是否进行生命体征检查:□是□□否 检查日期: |\_\_|\_|\_|-|\_\_|-|\_|-|\_(yyyy-mm-dd) 检查项目 检查结果 单位 临床意义 □正常 □异常无临床意义  $^{\circ}$ C 体温 □异常有临床意义 □未查 □正常 □异常无临床意义 脉搏 次/分 □异常有临床意义 □未查

次/分

□正常 □异常无临床意义

呼吸频率

| | | | □异常有临床意义 □未查 |
|---|---|---|---|
| | | | 71.11.14.11.11.11.11.11.11.11.11.11.11.11 |
| <br> 血压(收缩压) | mmHg | mmHg | □正常 □异常无临床意义 |
| | | □异常有临床意义 □未查 | |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 |
| III./II. (II.) (IV.II.) | | | □异常有临床意义 □未查 |
| | 四、 | 临床症状 | 犬 |
| 是否有新冠感染相关临床 | 症状:□是 [ | □否 | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | □呼吸短促或呼吸困难 □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 | □发热 □恶心 □呕吐 □腹泻 |
| │ □嗅觉减退 □味觉减退 | 艮 □其他症状 | : | |
| 开始日期: _ | - - | _ (уууу- | mm-dd) |
| 结束日期: | - - | _ (уууу- | mm-dd) |
| | 五、 | 体格检查 | 查 |
| 是否进行体格检查:□是 | □否 | | |
| 检查日期: | - - | _ (yyyy- | mm-dd) |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常□! | 异常无临床 | 意义 |
| AX IA VII | □异常有临床意 | 义 □ | 未查 |
| <br> 头颈部 | □正常 □! | 异常无临床 | 意义 |
| | □异常有临床意义 □未査 | | |
| 胸部 | □正常□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ | 异常无临床 | 意义 |
| 加加可 | □异常有临床意义 □未查 | | |
| 腹部 | □正常 □! | 异常无临床 | 意义 |
| 川文 口中 | □异常有临床意 | :义 □ | 未查 |
| 脊柱和四肢关节 | □正常 □! | 异常无临床 | 意义 |
| | □异常有临床意 | :义 □ | 未查 |
| 沖瓜 互 ひ | □正常□! | 异常无临床 | 意义 |
| 神经系统 | □异常有临床意 | :义 □ | 未查 |
| 皮肤 | □正常□! | 异常无临床 | 意义 |

| | □异常有临床意义 □未查 |
|---|---|
| 淋巴 | □正常 □异常无临床意义 |
| | □异常有临床意义 □未查 |
| 甘 (山 | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: mg | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnup | iravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ _ - - (yyyy-mm-dd) | |
| 是否持续: □是 □否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID | □TID □QW □PRN □其他 |
| 给药途径:□□服 □周 | |

| 注射 □其他 |
|-----------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称: □连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| <br> 初始给药日期: - - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|--------------------------------------------------------------|
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度 (FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药: □是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 □抗生素:□抗真菌类 □抗病毒类 |
| □糖皮质激素 |
| 日期: - - (yyyy-mm-dd)<br> 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: (vvvv-mm-dd) |

| 注:如有不良事件,请记录在"不良事件记录表" |
|---------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ _ - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型: □轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症: □是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ _ - - (yyyy-mm-dd) |
| 是否入院: □是 □否 |
| 入院日期: _ - _ - _ (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ - _ - _ (yyyy-mm-dd) |
| 是否出院: □是 □否 |
| 出院日期: _ - _ - _ (yyyy-mm-dd) |
| 是否死亡: □是 □否 |
| 死亡日期: _ - _ - _ (yyyy-mm-dd) |
| 死亡原因: |
#### 访视5-治疗期(第4天)

访视日期: |\_\_|\_|-|\_-|-|(yyyy-mm-dd) 一、新冠病毒核酸检测 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_\_|\_\_|-|\_\_|-|\_\_|-|(yyyy-mm-dd) 标本类型:□鼻咽拭子□□咽拭子 采样日期: |\_\_|\_|\_|-|\_\_|-|\_| (yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、血氧饱和度 是否进行血氧饱和度检查:□是□□否 检查日期: | | | | |-| | | (yyyy-mm-dd) 单位 检查项目 检查结果 临床意义 □正常 □异常无临床意义 指端脉氧饱和度 % □异常有临床意义 □未查 三、生命体征 是否进行生命体征检查:□是□□否 检查日期: |\_\_|\_|\_|-|\_\_|-|\_|-|\_(yyyy-mm-dd) 检查项目 检查结果 单位 临床意义 □正常 □异常无临床意义  $^{\circ}$ C 体温 □异常有临床意义 □未查 □正常 □异常无临床意义 脉搏 次/分 □异常有临床意义 □未查 呼吸频率 次/分 □正常 □异常无临床意义

| | | | □异常有临床意义 □未查 |
|---|---|---|---|
| 血压(收缩压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| | 四、 | 临床症状 | 比 |
| 是否有新冠感染相关临床 | 症状:□是 □ | □否 | |
| (如"是"),临床症状:[ | ]鼻塞或流涕 [ | □咽痛 □ | □呼吸短促或呼吸困难 □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 □ | □发热 □恶心 □呕吐 □腹泻 |
| □嗅觉减退 □味觉减退 | 艮 □其他症状 | : | |
| 开始日期: _ _ | - - | _ (yyyy- <u>1</u> | mm-dd) |
| 结束日期: _ | - _ - _ | _ (уууу- | mm-dd) |
| | 五、体格检查 | | |
| 是否进行体格检查:□是 □否 | | | |
| 检查日期: | - _ _ | _ (уууу-1 | mm-dd) |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常 □∮ | 异常无临床 | 意义 |
| ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | □异常有临床意 | :义 □ | 未查 |
| <b>头颈部</b> | □正常 □⅓ | 异常无临床 | 意义 |
| | □异常有临床意 | :义 🗆 | 未査 |
| 胸部 | □正常□⅓ | 异常无临床 | 意义 |
| ,,,,,,, | □异常有临床意 | 义 □ | 未查 |
| 腹部 | □正常 □⅓ | 异常无临床 | 意义 |
| )/文 Th | □异常有临床意 | :义 □ | 未查 |
| <br> 脊柱和四肢关节 | □正常 □! | 异常无临床 | 意义 |
| 日1111日放入 P | □异常有临床意 | :义 □ | 1未查 |
| 神经系统 | □正常 □! | | :意义 |
| 1世红尔坑 | □异常有临床意 | :义 □ | 未查 |
| 皮肤 | □正常 □! | 异常无临床 | 意义 |

| | □异常有临床意义 □未查 |
|---|---|
| NI err | □正常 □异常无临床意义 |
| 淋巴 | □异常有临床意义 □未查 |
| ++ /.L | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| <br> 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: mg | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnup | iravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ - _ - _ - _ (yyyy-mm-dd) | |
| 是否持续:□是□□否 | 是否持续: □是 □否 |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| <br> 给药剂量: _ m | g/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率:□QD□BID | □TID □QW □PRN □其他 |
| <br> 给药途径: □□服 □♬ | 引部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 □ |

| 注射 □其他 |
|-----------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|----------------------------------------------------------------|
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持:□是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药:□是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 □抗生素:□抗真菌类 □抗病毒类 |
| □糖皮质激素 |
| 日期: _ _ - - (yyyy-mm-dd)<br> 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 日期: |

| 注:如有不良事件,请记录在"不良事件记录表" |
|----------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - _ (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

# 访视 6-治疗期 (第5天)

| 访视日期: | _ | I | - | - | _ (yy | yy-mm-dd) |
|-------|---|---|---|---|--------|-----------|
|-------|---|---|---|---|--------|-----------|

| 一、新冠病毒核酸检测 | | | |
|--------------------------------|---------|----------|---------------|
| 是否进行新冠病毒核酸检测: | □是□□酉 | ; | |
| 检测日期: - | - | (yyyy-mm | ı–dd) |
| 标本类型:□鼻咽拭子□□ | 口咽拭子 | | |
| 采样日期: _ _ - | - | (yyyy-mm | i–dd) |
| 新型冠状病毒 ORF1ab 基因: | □阴性 □ | 阳性 | |
| 新型冠状病毒 ORF1ab 基因 Ct | 值: | _ | |
| 新型冠状病毒 N 基因: □阴性 | □阳性 | | |
| 新型冠状病毒 N 基因 Ct 值: | | | |
| | 二、胸部 | 部影像学检 | :测* |
| 是否进行胸部影像学检查:□ | ]是 口否 | ; | |
| 检查日期: _ _ _ - | | | |
| 检查名称 检查内容 临床意义 | | | |
| 胸部(肺部)CT | | | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 胸部(肺部)X射线 | | | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| | 三、 | 血氧饱和度 | Ē |
| 是否进行血氧饱和度检查:□是 □否 | | | |
| 检查日期: _ - - (yyyy-mm-dd) | | | |
| 检查项目 检查 | <b></b> | 单位 | 临床意义 |
| <br> <br> 指端脉氧饱和度 | | 0' | □正常 □异常无临床意义 |
| 7日州加平、地平/交 | | % | □异常有临床意义 □未查 |
| 四、生命体征 | | | |

| 是否进行生命体征检查: | □是 □否 | | |
|---|---|---|---|
| 检查日期: _ - _ - _ - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 体温 | | $^{\circ}$ | □正常 □异常无临床意义 |
| 744皿 | | C | □异常有临床意义 □未查 |
| <br> 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| 744-4-4 | | 0,4,74 | □异常有临床意义 □未查 |
| 呼吸频率 | | 次/分 | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| <br> 血压(收缩压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| <br> 血压(舒张压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 五、临床症状 | | | |
| 是否有新冠感染相关临床症状:□是 □否 | | | |
| (如"是"),临床症状:□鼻塞或流涕 □咽痛 □呼吸短促或呼吸困难 □咳嗽 □ | | | |
| <br> 乏力 □肌肉或身体痛 □头痛 □寒战 □发热 □恶心 □呕吐 □腹泻 | | | |
| □嗅觉减退 □味觉减退 □其他症状: | | | |
| <br> 开始日期 <b>:</b> _ _ _ | - _ - _ | _ (yyyy- <u>r</u> | nm-dd) |
| <br> 结束日期: _ _ _ | - _ _ | _ (yyyy-r | nm-dd) |
| | 六、 | 体格检查 | <u> </u> |
| 是否进行体格检查:□是 | □否 | | |
| 检查日期: _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常 □∮ | 异常无临床 | 意义 |
| 74X 173 Vu | □异常有临床意 | 义 口 | 未查 |
| 头颈部<br>头颈部 | □正常 □∮ | 异常无临床 | 意义 |
| | □异常有临床意 | 义 口 | 未查 |
| 胸部 | □正常 □∮ | 异常无临床 | 意义 |
| 시는 10년(N | □异常有临床意 | 义 口 | 未查 |

| IV는 것만 | □正常 □ | ]异常无临床 | 意义 | |
|---|---|---|---|---|
| 腹部 | □异常有临床 | 意义 □ | 未查 | |
| 脊柱和四肢关节 | □正常 □ | ]异常无临床 | 意义 | |
| 有性和四版大 | □异常有临床 | 意义 □ | 未查 | |
| 神经系统 | □正常 □ | ]异常无临床 | 意义 | |
| | □异常有临床 | 意义 □ | 未查 | |
| 皮肤 | □正常 □ | □正常 □异常无临床意义 | | |
| /X/IX | □异常有临床 | □异常有临床意义 □未查 | | |
| 淋巴 | □正常 □ | ]异常无临床 | 意义 | |
| 7/T L | □异常有临床 | 意义 □ | 未查 | |
| 其他 | □正常 □ | ]异常无临床 | 意义 | |
| 光吧 | □异常有临床 | 意义 □ | 未查 | |
| 七、实验室检查 | | | | |
| 是否进行血常规检查:□是 □否 | | | | |
| 检查日期: - - (yyyy-mm-dd) | | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 | |
| 红细胞计数 (RBC) | | $10^{12}/{ m L}$ | □正常 □异常无临床意义 | |
| 红细胞计数(NDC) | | 1012/L | □异常有临床意义 □未查 | |
| 白细胞计数(WBC) | | | | _ |
| 四細胞( 数(wbc) | | 109/I | □正常 □异常无临床意义 | |
| | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 □异常有临床意义 □未查 | |
| 血红蛋白(Hb) | | | | |
| 血红蛋白(Hb) | | 10 <sup>9</sup> /L<br>g/L | □异常有临床意义 □未查 | |
| | | g/L | □异常有临床意义 □未查<br>□正常 □异常无临床意义 | _ |
| 血红蛋白(Hb)<br>血小板计数(PLT) | | | □异常有临床意义 □未查 □正常 □异常无临床意义 □异常有临床意义 □未查 | |
| 血小板计数(PLT) | | g/L<br>10 <sup>9</sup> /L | <ul><li>□ 异常有临床意义</li><li>□ 正常</li><li>□ 异常无临床意义</li><li>□ □ 异常有临床意义</li><li>□ 正常</li><li>□ 异常无临床意义</li></ul> | |
| | | g/L | <ul><li>□ 异常有临床意义</li><li>□ 正常</li><li>□ 异常无临床意义</li><li>□ □ 异常无临床意义</li><li>□ 正常</li><li>□ 异常无临床意义</li><li>□ □ 异常无临床意义</li><li>□ 异常有临床意义</li><li>□ □ 未查</li></ul> | |
| 血小板计数(PLT) | | g/L<br>10 <sup>9</sup> /L | □ 异常有临床意义 □ 未查 □ 正常 □ 异常无临床意义 □ 正常 □ 异常无临床意义 □ 异常有临床意义 □ 未查 □ 正常 □ 异常无临床意义 □ 正常 □ 异常无临床意义 | |

| ₩ III ₩ ₩ ( I ) | 109/ | | □正常 □异常无临床意义 |
|-----------------------|------|--------------------|---------------|
| 淋巴细胞计数(Lym) | | 10 <sup>9</sup> /L | □异常有临床意义 □未查 |
| 是否进行血生化检查: □ | 是□否 | | |
| 检查日期: | - - | (yyyy-r | nm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| | | □U/L | □正常 □异常无临床意义 |
| 谷丙转氨酶(ALT) | | □IU/L | □异常有临床意义 □未查 |
| ◇ 古 杜 与 ■ | | U/L | □正常 □异常无临床意义 |
| 谷草转氨酶(AST) | | □IU/L | □异常有临床意义 □未查 |
| 石矿。44. 五米 亚公 亚尔(AI D) | | U/L | □正常 □异常无临床意义 |
| 碱性磷酸酶(ALP) | | □IU/L | □异常有临床意义 □未查 |
| 总胆红素 (STB) | | □umo1/L | □正常 □异常无临床意义 |
| 心胆红系 (SID) | | □mg/d1 | □异常有临床意义 □未查 |
| 古体阳尔圭(NDII) | | □umo1/L | □正常 □异常无临床意义 |
| 直接胆红素(DBIL) | | □mg/d1 | □异常有临床意义 □未查 |
| 总蛋白(TP) | | g/L | □正常 □异常无临床意义 |
| | | 0, - | □异常有临床意义 □未查 |
| 白蛋白(ALB) | | g/L | □正常 □异常无临床意义 |
| | | O, | □异常有临床意义 □未查 |
| 尿素氮(BUN) | | mmo1/L | □正常 □异常无临床意义 |
| MAN AN (BOTT) | | mmo 17 E | □异常有临床意义 □未查 |
| 血肌酐(Cr) | | □mg/d1 | □正常 □异常无临床意义 |
| (急性肾衰□是 □否) | | □umo1/L | □异常有临床意义 □未查 |
| 血糖(Glu) | | mmo1/L | □正常 □异常无临床意义 |
| IIIL7/档(GIU) | | IIIIIO1/L | □异常有临床意义 □未查 |
| 尿酸(UA) | | μ mol/L | □正常 □异常无临床意义 |
| /水質(UA) | | h IIIOI/L | □异常有临床意义 □未查 |

| <i>Н</i> Ш (177) | | mm o 1 /I | □正常 □异常无临床意义 |
|---------------------------|--------|---------------------|------------------|
| 钾(K) | | mmo1/L | □异常有临床意义 □未查 |
| 钠 (Na) | | mmo1/L | □正常 □异常无临床意义 |
| ty (Na) | | MMO1/L | □异常有临床意义 □未查 |
| 复(01) | | 1 /1 | □正常 □异常无临床意义 |
| 氯 (C1) | | mmo1/L | □异常有临床意义 □未查 |
| 是否进行凝血功能检查: | □是 □否 | | |
| 检查日期: | - - | (уууу-г | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 海南南百叶词 (DT) | | _ | □正常 □异常无临床意义 |
| 凝血酶原时间(PT) | | S | □异常有临床意义 □未查 |
| 活化部分凝血活酶时间 | | _ | □正常 □异常无临床意义 |
| (APTT) | | S | □异常有临床意义 □未查 |
| | | □g/L | □正常 □异常无临床意义 |
| 纤维蛋白原(Fg) | | □mg/d1 | □异常有临床意义 □未查 |
| 생조 do 표는 마나 라크 (''''''' \ | | | □正常 □异常无临床意义 |
| 凝血酶时间(TT) | | S | □异常有临床意义 □未查 |
| n 一取从(n n: .) | | □ µ g/L | □正常 □异常无临床意义 |
| D-二聚体(D-Dimer) | | □mg/L | □异常有临床意义 □未查 |
| 是否进行动脉血气分析检 | 测:□是 □ | ]否 | |
| 检查日期: _ | - - _ | (yyyy- <sub>1</sub> | mm-dd) |
| 检查项目 | 检查结果 | 単位 | 临床意义 |
| РН | | | □正常 □异常无临床意义 |
| 111 | | | □异常有临床意义 □未查 |
| 血氧饱和度 | | % | □正常 □异常无临床意义 |
| ,, =,, 2, | | | □异常有临床意义 □未查 |
| <br>二氧化碳分压(PaCO₂) | | mmHg | □正常 □异常无临床意义 |
| - | | | □异常有临床意义 □未查 |
| 氧分压 (PaO <sub>2</sub> ) | | mmHg | □正常 □异常无临床意义 □未杳 |

| 碳酸氢(HCO3¯) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
|---|---|---|---|
| 氧合指数(PaO <sub>2</sub> /FiO <sub>2</sub> ) | | mmHg | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 是否进行血脂检测:□是 | <br>□否 | 1 | |
| <br> 检查日期: | - _ - | (уууу- | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 总胆固醇 (TC) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 甘油三酯(TG) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 高密度脂蛋白(HDL-C) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 低密度脂蛋白(LDL-C) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| | 八、 | 炎症标志 | 物 |
| 是否进行炎症标志物检查:□是 □否 | | | |
| 检查日期: | - - | (yyyy- | mm-dd) |
| 检查项目 | 检查结果 | 単位 | 临床意义 |
| | | □ µ g/L | |
| C 反应蛋白 | | □mg/d1 | □正常 □异常无临床意义<br> □异常有临床意义 □未查 |
| | | □mg/L | |
| 降钙素原 | | ng/ml | □正常 □异常无临床意义 |
| 叶小水小 | | 118/ 1111 | □异常有临床意义 □未查 |
| 九、治疗方案 | | | |
| 新冠感染药物治疗 | | | |
| 来瑞特韦给药情况 | | | |
| 药物规格: mg | | | |
| 初始给药日期: _ - _ - _ - _ (yyyy-mm-dd) | | | |
| 是否持续: □是 □否 | | | |
| 结束给药日期: - - - (yyyy-mm-dd) | | | |
| 给药剂量: mg | | | |

| 给药频率: □QD □BID □TID □QW □PRN □其他 |
|-------------------------------------------------------|
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg |
| 其他新冠治疗药物给药情况 |
| <br> 抗病毒小分子药物 |
| │<br> 药物名称: □奈玛特韦片/利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |

| 中和抗体 |
|---|
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物注射 □其他 |
| <br> 注射 □其他 |
| 注射 □其他<br>总剂量: mg 或 g |
| 注射 □其他<br>总剂量: mg 或 g<br><b>新冠非药物干预:</b> |
| 注射 □其他<br>总剂量: mg 或 g<br><b>新冠非药物干预:</b><br>抗凝治疗: □是 □否 |
| 注射 □其他<br>总剂量: mg 或 g<br>新冠非药物干预:<br>抗凝治疗: □是 □否<br>如"是"请勾选: □低分子肝素 □普通肝素 □其他 |

| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(Fi02): %; 小时/天; |
|--------------------------------------------------------|
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 十、合并用药 |
| 是否发生合并用药:□是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 |
| □抗生素: □抗真菌类 □抗病毒类 |
| □糖皮质激素 |
| 日期: - - (yyyy-mm-dd) 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 十一、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: - - (yyyy-mm-dd) |
| 注: 如有不良事件,请记录在"不良事件记录表" |
| 十二、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: - - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ - - (yyyy-mm-dd) |
| 入院科室: |

| 是否进入 ICU: □是 □否 |
|---------------------------------|
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |
| 十三、新冠病毒基因检测 |
| 是否保留受试者新冠病毒核酸检测样本: □是 □否 |
| 标本类型:□鼻拭子 □咽拭子 |

### 访视7-治疗期(第6天)

| 访视日期: _ _ - _ - _ - (yyyy-mm-dd) | | | |
|---|---|---|---|
| | 一、新冠 | 病毒核酢 | <b>发检测</b> |
| 是否进行新冠病毒植 | 亥酸检测:□是□□否 | | |
| 检测日期: _ | _ - - | (yyyy- <sub>l</sub> | mm-dd) |
| 标本类型:□鼻咽拮 | 式子 □□咽拭子 | | |
| <br> 采样日期: _ | _ - - | (уууу- | mm-dd) |
| 新型冠状病毒 ORF1a | ab 基因: □阴性 □阝 | 阳性 | |
| 新型冠状病毒 ORF1a | ab 基因 Ct 值: | - | |
| 新型冠状病毒 N 基团 | 因:□阴性 □阳性 | | |
| │<br>│新型冠状病毒 N 基团 | 因 Ct 值: | | |
| 二、血氧饱和度 | | | |
| 是否进行血氧饱和原 | 度检查:□是□□否 | | |
| 检查日期: _ | _ - - | (уууу- | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 指端脉氧饱和度 | | % | □正常 □异常无临床意义 |
| 1日圳脉苇、地和皮 | | 70 | □异常有临床意义 □未查 |
| 三、生命体征 | | | |
| 是否进行生命体征检查:□是 □否 | | | |
| 检查日期: _ _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 体温 | | $^{\circ}$ | □正常 □异常无临床意义 |
| , | | | □异常有临床意义 □未查 |
| <br> 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |

次/分

呼吸频率

□正常

□异常无临床意义

| | | | □异常有□ | 临床意义 | □未查 |
|---|---|---|---|---|---|
| 加压 ()协统压) | 血压(收缩压) mmHg | mmUa | □正常 | □异常无 | 临床意义 |
| 皿压 (収細压) | | □异常有□ | 临床意义 | □未查 | |
| 血压(舒张压) mmHg | mmHg | □正常 | □异常无 | 临床意义 | |
| шиле (на јуле) | | | □异常有□ | 临床意义 | □未查 |
| 四、临床症状 | | | | | |
| 是否有新冠感染相关临床症状:□是 □否 | | | | | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | □呼吸短促耳 | <b></b> | □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 | □发热 □ | ]恶心 □ | 呕吐 □腹泻 |
| │ □嗅觉减退 □味觉减退 | 艮 □其他症状 | : | | | |
| <br> 开始日期: _ _ | - - | _ (уууу- | mm-dd) | | |
| 结束日期: _ _ | - - | _ (уууу- | mm-dd) | | |
| | 五、 | 体格检查 | 生 | | |
| 是否进行体格检查:□是 | □否 | | | | |
| 检查日期: _ _ | - - | _ (уууу- | mm-dd) | | |
| 检查项目 | 临 | 床意义 | | 若有异 | 常,请描述 |
| 一般情况 | □正常 □∮ | 异常无临床 | 意义 | | |
| /2X 113 / U | □异常有临床意 | :义 □ | 未查 | | |
| | □正常□⅓ | | | | |
| | □异常有临床意 | | | | |
| <br> 胸部 | □正常□፵ | 异常无临床 | 意义 | | |
| | □异常有临床意 | 义 □ | 未查 | | |
| 腹部 | □正常 □! | 异常无临床 | 意义 | | |
| VS ロP | □异常有临床意 | 义 □ | 未查 | | |
| 26 L2 7nm 1L V. ++ | □正常 □∮ | 异常无临床 | 意义 | | |
| 骨柱和四肢关节<br> | □异常有临床意 | :义 □ | 未查 | | |
| 油が だか | □正常 □⅓ | 异常无临床 | 意义 | | |
| 神经系统 | □异常有临床意 | :义 □ | 未查 | | |
| 皮肤 | □正常 □┆ | 异常无临床 | 意义 | | |

| | □异常有临床意义 □未查 |
|---|---|
| NI err | □正常 □异常无临床意义 |
| 淋巴 | □异常有临床意义 □未查 |
| | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| <br> 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: _ mg | |
| 给药频率:□QD □BID | □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnup | iravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 | _ |
| 药物规格: mg 或 g | |
| 初始给药日期: _ - - (yyyy-mm-dd) | |
| 是否持续: □是 □否 | |
| 结束给药日期: _ - - (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| <br> 给药途径: □□服 □♬ | 引部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 □ |

| 注射 □其他 |
|-----------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|---|
| <br> 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持:□是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药:□是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 □抗生素:□抗真菌类 □抗病毒类 |
| □糖皮质激素 |
| 日期: _ _ - - - (yyyy-mm-dd)<br> 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 日期: |

| 注:如有不良事件,请记录在"不良事件记录表" |
|----------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - _ (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

# 访视8-治疗期(第7天)

| 访视日期: - - - (yyyy-mm-dd) | | | | |
|---|---|---|---|---|
| 一、新冠病毒核酸检测 | | | | |
| 是否进行新冠病毒核 | 酸检测:□是□□否 | ; | | |
| 检测日期: _ | _ _ - - | (yyyy-mm | ı–dd) | |
| 标本类型:□鼻咽拭 | 子 口口咽拭子 | | | |
| <br> 采样日期: _ | _ _ - - _ | (yyyy-mm | ı–dd) | |
| 新型冠状病毒 ORF1ab | 基因:□阴性 □ | 阳性 | | |
| 新型冠状病毒 ORF1ab | 基因 Ct 值: | | | |
| 新型冠状病毒 N 基因: | :□阴性 □阳性 | | | |
| 新型冠状病毒 N 基因 | Ct 值: | | | |
| | 二、血氧饱和度 | | | |
| 是否进行血氧饱和度 | 是否进行血氧饱和度检查: □是 □否 | | | |
| 检查日期: - - (yyyy-mm-dd) | | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 | |
| 指端脉氧饱和度 | | % | □正常 □异常尹 | <b>尼临床意义</b> |
| 1日 圳 / 斯 / 11 / 12 / 12 / 12 / 12 / 12 / 12 | | 70 | □异常有临床意义 | □未查 |
| 三、生命体征 | | | | |
| 是否进行生命体征检查:□是 □否 | | | | |
| 检查日期: _ _ - - (yyyy-mm-dd) | | | | |

| 检查项目 | 检查结果 | 单位 | 临床意义 |
|-------|------|------------|---------------|
| 体温 | | $^{\circ}$ | □正常 □异常无临床意义 |
| r+ um | | | □异常有临床意义 □未查 |
| 脉搏 | 次/分 | | □正常 □异常无临床意义 |
| | | 10(7)) | □异常有临床意义 □未查 |
| 呼吸频率 | | 次/分 | □正常 □异常无临床意义 |
| | | (A) | □异常有临床意义 □未查 |

| 血压(收缩压) | | mmHg | □正常 | □异常无临 | 床意义 |
|---|---|---|---|---|---|
| III./II. \ \\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 8 | □异常有□ | 临床意义 | □未查 | |
| 血压(舒张压) | | mmHg | | □异常无临 | |
| | | | □异常有□ | 临床意义 | □未査 |
| | 四、 | 临床症状 | 7 | | |
| 是否有新冠感染相关临床 | 症状:□是□ | □否 | | | |
| (如"是"),临床症状:□鼻塞或流涕 □咽痛 □呼吸短促或呼吸困难 □咳嗽 □ | | | | | □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 □ | 〕发热 □ | ]恶心 □呕 | 吐 □腹泻 |
| □嗅觉减退 □味觉减过 | 艮 □其他症状 | : | | | |
| 开始日期: _ _ | - - | _ (yyyy- <u>r</u> | nm-dd) | | |
| 结束日期: _ | - _ - _ | _ (yyyy-r | nm-dd) | | |
| | 五、 | 体格检查 | <u> </u> | | |
| 是否进行体格检查:□是 | □否 | | | | |
| 检查日期: _ _ | - _ - _ | _ (yyyy-r | nm-dd) | | |
| 检查项目 | 临床意义 若有异常,请描述 | | | ,请描述 | |
| 一般情况 | □正常 □异常无临床意义 | | | | |
| /2/113/24 | □异常有临床意 | 义 口: | 未查 | | |
| | □正常 □∮ | 异常无临床 | 意义 | | |
| 2 | □异常有临床意 | 义 口: | 未查 | | |
| 胸部 | □正常 □∮ | 异常无临床 | 意义 | | |
| 月岡 青13 | | | | | |
| | □异常有临床意 | 义 口: | 未查 | | |
| FG か7 | □异常有临床意<br>□正常 □5 | | | | |
| 腹部 | | 异常无临床: | 意义 | | |
| | □正常 □∮ | 异常无临床: | 意义<br>未查 | | |
| 腹部 | □正常 □昇常有临床意 | 异常无临床<br>:义 □<br>异常无临床 | 意义 未查 意义 | | |
| 脊柱和四肢关节 | □正常 □ | 异常无临床<br>: 义 □ | 意义<br>未查<br>意义<br>未查 | | |
| | □正常 □昇常有临床意<br>□正常 □昇<br>□异常有临床意 | 异常无临床<br>:义 □<br>异常无临床<br>:义 □<br>异常无临床 | 意义<br>未查<br>意义<br>未查<br>意义 | | |
| 脊柱和四肢关节 | □正常 □射 □异常有临床意 □正常 □射 □异常有临床意 □正常 □引 | 异常无临床<br>: 义 □ | 意义<br>未 意<br>意 在<br>意 文<br>未 意<br>未 意 | | |

| 34 III | □正常 □异常无临床意义 |
|---|---|
| 淋巴 | □异常有临床意义 □未查 |
| ++- /-1. | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: _ mg | |
| 给药频率:□QD □BID | □TID □QW □PRN □其他 |
| 给药途径:□□服 □原 | 局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 | |
| 总剂量: _ mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnup | iravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ - _ - _ (yyyy-mm-dd) | |
| 是否持续: □是 □否 | |
| 结束给药日期: _ - _ - _ - _ (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |

| 总剂量: mg 或 g |
|-----------------------------------------|
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |

| 结束给药日期: _ - _ - _ (yyyy-mm-dd) |
|-------------------------------------------------|
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持:□是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃;吸氧浓度(Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药:□是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物: □多巴胺 □肾上腺素 □去甲肾上腺素 □ |
| □抗生素: □抗真菌类 □抗病毒类 □糖皮质激素 |
| 日期: _ - - (yyyy-mm-dd) |
| 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 是否发生安全性事件: □是 □否 |
| 日期: _ _ - - (yyyy-mm-dd) |
| 注: 如有不良事件,请记录在"不良事件记录表" |

| 九、疾病诊断信息 |
|--------------------------------|
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: - - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: - - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: - - - (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: - - - (yyyy-mm-dd) |
| 死亡原因: |

#### 访视9-治疗期(第8天)

访视日期: |\_\_|\_|-|\_-|-|(yyyy-mm-dd) 一、新冠病毒核酸检测 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_\_|\_\_|-|\_\_|-|\_\_|-|(yyyy-mm-dd) 标本类型:□鼻咽拭子□□咽拭子 采样日期: |\_\_|\_|\_|-|\_\_|-|\_|-|(yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、血氧饱和度 是否进行血氧饱和度检查:□是□□否 检查日期: | | | | |-| | | (yyyy-mm-dd) 单位 检查项目 检查结果 临床意义 □正常 □异常无临床意义 指端脉氧饱和度 % □异常有临床意义 □未查 三、生命体征 是否进行生命体征检查:□是□□否 检查日期: |\_\_|\_|\_|-|\_\_|-|\_|-|\_(yyyy-mm-dd) 检查项目 检查结果 单位 临床意义 □正常 □异常无临床意义  $^{\circ}$ C 体温 □异常有临床意义 □未查 □正常 □异常无临床意义 次/分 脉搏 □异常有临床意义 □未查 呼吸频率 次/分 □正常 □异常无临床意义

| | | | □异常有临床意义 □未查 |
|---|---|---|---|
| | | | 71.11.14.11.11.11.11.11.11.11.11.11.11.11 |
| <br> 血压(收缩压) | mmHg | mmHg | □正常 □异常无临床意义 |
| mayar ( DV-)H/LL / | | | □异常有临床意义 □未查 |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 四、临床症状 | | | |
| 是否有新冠感染相关临床症状: □是 □否 | | | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | □呼吸短促或呼吸困难 □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 | □发热 □恶心 □呕吐 □腹泻 |
| │ □嗅觉减退 □味觉减退 | 艮 □其他症状 | : | |
| 开始日期: _ | - - | _ (уууу- | mm-dd) |
| 结束日期: | - - | _ (уууу- | mm-dd) |
| | 五、 | 体格检查 | 查 |
| 是否进行体格检查:□是 | □否 | | |
| 检查日期: | - - | _ (yyyy- | mm-dd) |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常□! | 异常无临床 | 意义 |
| AX IA VII | □异常有临床意义 □未査 | | |
| <br> 头颈部 | □正常 □! | 异常无临床 | 意义 |
| | □异常有临床意 | 义 □ | 未查 |
| 胸部 | □正常□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ | 异常无临床 | 意义 |
| □ | □异常有临床意义 □未查 | | |
| I/드 수대 | □正常 □! | 异常无临床 | 意义 |
| 腹部 | □异常有临床意 | :义 □ | 未查 |
| ₩ 15 10 mm u+ W ++ | □正常 □! | 异常无临床 | 意义 |
| 脊柱和四肢关节 | □异常有临床意 | :义 □ | 未查 |
| 沖瓜 互 ひ | □正常□! | 异常无临床 | 意义 |
| 神经系统 | □异常有临床意 | :义 □ | 未查 |
| 皮肤 | □正常 □! | 异常无临床 | 意义 |

| | □异常有临床意义 □未查 |
|---|---|
| NI err | □正常 □异常无临床意义 |
| 淋巴 | □异常有临床意义 □未查 |
| | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| <br> 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: _ mg | |
| 给药频率:□QD □BID | □TID □QW □PRN □其他 |
| 给药途径:□□服 □原 | 引部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称: □奈玛特韦片/利托那韦片 (Paxlovid) □先诺特韦片/利托那韦片 (先诺欣) | |
| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 | |
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ _ - - (yyyy-mm-dd) | |
| 是否持续: □是 □否 | |
| 结束给药日期: _ - - (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| <br> 给药途径: □□服 □♬ | 引部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 □ |

| 注射 □其他 |
|------------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称:□COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| <br> 初始给药日期: _ _ - - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|-------------------------------------------------|
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药: □是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 |
| □抗生素: □抗真菌类 □抗病毒类 □糖皮质激素 |
| 日期: - - (yyyy-mm-dd) |
| 注:如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: - - (yyyy-mm-dd) |

| 注: 如有不良事件,请记录在"不良事件记录表" |
|----------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - _ (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

### 访视10-治疗期(第9天)

访视日期: |\_\_|\_|-|\_-|-|(yyyy-mm-dd) 一、新冠病毒核酸检测 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_\_|\_\_|-|\_\_|-|\_\_|-|(yyyy-mm-dd) 标本类型:□鼻咽拭子□□咽拭子 采样日期: |\_\_|\_|\_|-|\_\_|-|\_|-|(yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、血氧饱和度 是否进行血氧饱和度检查:□是□□否 检查日期: | | | | |-| | | (yyyy-mm-dd) 单位 检查项目 检查结果 临床意义 □正常 □异常无临床意义 指端脉氧饱和度 % □异常有临床意义 □未查 三、生命体征 是否进行生命体征检查:□是□□否 检查日期: |\_\_|\_|\_|-|\_\_|-|\_|-|\_(yyyy-mm-dd) 检查项目 检查结果 单位 临床意义 □正常 □异常无临床意义  $^{\circ}$ C 体温 □异常有临床意义 □未查 □正常 □异常无临床意义 脉搏 次/分 □异常有临床意义 □未查

次/分

□正常 □异常无临床意义

呼吸频率

| | | | □异常有临床意义 □未查 | |
|---|---|---|---|--|
| | | | 71.11.14.11.11.11.11.11.11.11.11.11.11.11 | |
| <br> 血压(收缩压) | mmHg | mmHg | □正常 □异常无临床意义 | |
| mayar ( DV-)H/LL / | | | □异常有临床意义 □未查 | |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 | |
| | | | □异常有临床意义 □未查 | |
| 四、临床症状 | | | | |
| 是否有新冠感染相关临床症状: □是 □否 | | | | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | □呼吸短促或呼吸困难 □咳嗽 □ | |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 | □发热 □恶心 □呕吐 □腹泻 | |
| │ □嗅觉减退 □味觉减退 | 艮 □其他症状 | : | | |
| 开始日期: _ | - - | _ (уууу- | mm-dd) | |
| 结束日期: | - - | _ (уууу- | mm-dd) | |
| | 五、 | 体格检查 | 查 | |
| 是否进行体格检查:□是 | □否 | | | |
| 检查日期: | - - | _ (yyyy- | mm-dd) | |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 | |
| 一般情况 | □正常□! | 异常无临床 | 意义 | |
| AX IA VII | □异常有临床意义 □未査 | | | |
| <br> 头颈部 | □正常 □! | 异常无临床 | 意义 | |
| | □异常有临床意 | 义 □ | 未查 | |
| 胸部 | □正常□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ | 异常无临床 | 意义 | |
| □ | □异常有临床意义 □未查 | | | |
| I/드 수대 | □正常 □! | 异常无临床 | 意义 | |
| 腹部 | □异常有临床意 | :义 □ | 未查 | |
| ₩ 15 10 mm u+ W ++ | □正常 □! | 异常无临床 | 意义 | |
| 脊柱和四肢关节 | □异常有临床意 | :义 □ | 未查 | |
| 沖瓜 互 ひ | □正常□! | 异常无临床 | 意义 | |
| 神经系统 | □异常有临床意 | :义 □ | 未查 | |
| 皮肤 | □正常□! | 异常无临床 | 意义 | |
| | □异常有临床意义 □未查 |
|----------------|------------------------------------|
| NI FF | □正常 □异常无临床意义 |
| 淋巴 | □异常有临床意义 □未查 |
| # 14 | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 六、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| 药物规格: _ mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: _ mg | |
| 给药频率:□QD □BID | □TID □QW □PRN □其他 |
| 给药途径:□□服 □周 | 局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnup | iravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 | _ |
| 药物规格: _ mg | 或g |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是□□否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: _ m | g/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率:□QD □BID | □TID □QW □PRN □其他 |
| 给药途径:□□服 □周 | 局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |

| 注射 □其他 |
|-----------------------------------------|
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称: □连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| <br> 初始给药日期: - - - (yyyy-mm-dd) |

| 是否持续: □是 □否 |
|-------------------------------------------------|
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 七、合并用药 |
| 是否发生合并用药: □是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 |
| □抗生素: □抗真菌类 □抗病毒类 □糖皮质激素 |
| 日期: _ - - (yyyy-mm-dd) |
| 注:如有合并用药,详细用药请记录在"合并用药记录表" |
| 八、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: - - (yyyy-mm-dd) |

| 注: 如有不良事件,请记录在"不良事件记录表" |
|----------------------------------|
| 九、疾病诊断信息 |
| 是否确诊新型冠状病毒感染: □是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

#### 访视 11-治疗期 (第 10 天)

访视日期: |\_\_|\_|-|\_\_|-|\_| (yyyy-mm-dd) 一、新冠病毒核酸检测 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_\_|\_\_|-|\_\_|-|\_\_| (yyyy-mm-dd) 标本类型:□鼻咽拭子 □□咽拭子 采样日期: | | | | |-| | | (yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、胸部影像学检测\* 是否进行胸部影像学检查:□是□□否 检查日期: |\_\_|\_|\_|-|\_\_|-|\_\_| (yyyy-mm-dd) 检查名称 检查内容 临床意义 胸部(肺部)CT □正常 □异常无临床意义 □异常有临床意义 □未查 胸部 (肺部) X 射线 □正常 □异常无临床意义 □异常有临床意义 □未查 三、血氧饱和度 是否进行血氧饱和度检查:□是□□否 检查日期: | (yyyy-mm-dd) 检查项目 单位 临床意义 检查结果 □正常 □异常无临床意义 指端脉氧饱和度 % □异常有临床意义 □未查

四、生命体征

| 是否进行生命体征检查: | □是 □否 | | |
|---|---|---|---|
| 检查日期: _ _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 体温 | | °C | □正常 □异常无临床意义 |
| (本) | | C | □异常有临床意义 □未查 |
| 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| )N/144 | | | □异常有临床意义 □未查 |
| 呼吸频率 | | 次/分 | □正常 □异常无临床意义 |
| 3 /2// 1 | | | □异常有临床意义 □未查 |
| 血压(收缩压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| 血压(舒张压) | | mmHg | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查 |
| | 五、 | 临床症状 | F |
| 是否有新冠感染相关临床 | 症状:□是□□ | ]否 | |
| (如"是"),临床症状:□鼻塞或流涕 □咽痛 □呼吸短促或呼吸困难 □咳嗽 □ | | | |
| 乏力 □肌肉或身体痛 □头痛 □寒战 □发热 □恶心 □呕吐 □腹泻 | | | |
| □嗅觉减退 □味觉减退 □其他症状: | | | |
| <br>开始日期: _ - - - (yyyy-mm-dd) | | | |
| 结束日期: _ - - (yyyy-mm-dd) | | | |
| 六、体格检查 | | | |
| 是否进行体格检查:□是 | □否 | | |
| 检查日期: _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常 □∮ | 异常无临床 | 意义 |
| 74411792 | □异常有临床意 | 义 口: | 未查 |
| 头颈部 | □正常 □∮ | 早常无临床: | 意义 |
| | □异常有临床意 | 义 口: | 未查 |
| 胸部 | □正常 □∮ | 早常无临床: | 意义 |
| 別的 守り | □异常有临床意 | 义 口: | 未查 |

| DC 50 | □正常 □ | ]异常无临床 | 意义 | | |
|---|---|---|---|---|---|
| 腹部 | □异常有临床 | 意义 □ | 未查 | | |
| <b>炎</b> 比和Ⅲ肚子芸 | □正常 □ | ]异常无临床 | 意义 | | |
| 骨柱和四肢关节<br> | □异常有临床 | 意义 □ | 未查 | | |
| 神经系统 | □正常 □ | ]异常无临床 | 意义 | | |
| 押 | □异常有临床 | 意义 □ | 未查 | | |
| 皮肤 | □正常 □ | 〕异常无临床 | 意义 | | |
| /文/AX | □异常有临床 | 意义 □ | 未查 | | |
| 淋巴 | □正常 □ | 〕异常无临床 | 意义 | | |
| 71T L | □异常有临床 | 意义 □ | 未查 | | |
| 其他 | □正常 □ | 〕异常无临床 | 意义 | | |
| <b>共</b> 他 | □异常有临床 | 意义 □ | 未查 | | |
| | 七、 | 实验室检 | 查# | | |
| 是否进行血常规检查:□ | 是□否 | | | | |
| <br> 检查日期: | _ - - | (yyyy- | nm-dd) | | |
| 检查日期: <br>检查项目 | - - _ | (yyyy-<br> <br> 单位 | | 临床意》 | Z. |
| 检查项目 | | 单位 | | | |
| | | | I | ]异常无 | 临床意义 |
| 检查项目<br>红细胞计数(RBC) | | 单位<br>10 <sup>12</sup> /L | □正常 □ | ]异常无<br>意义 | 临床意义<br>□未査 |
| 检查项目 | | 单位 | □正常 □ | | 临床意义<br>□未査<br>临床意义 |
| 检查项目 红细胞计数(RBC) 白细胞计数(WBC) | | 单位<br>10 <sup>12</sup> /L<br>10 <sup>9</sup> /L | □正常□□正常□□正常□□□正常□□□□□□□□□□□□□□□□□□□□□□ | 意义 异常无意义 | 临床意义 □未查 临床意义 □未查 |
| 检查项目<br>红细胞计数(RBC) | | 单位<br>10 <sup>12</sup> /L | □正常 □<br>□异常有临床;<br>□正常 □<br>□异常有临床; | ]异常无<br>意义<br>]异常无<br>意义<br>]异常无 | 临床意义<br>□未查<br>临床意义<br>□未查<br>临床意义 |
| 检查项目 红细胞计数(RBC) 白细胞计数(WBC) 血红蛋白(Hb) | | 单位<br>10 <sup>12</sup> /L<br>10 <sup>9</sup> /L<br>g/L | □正常 □ | 意义<br>]异常无<br>意义<br>]异常无<br>意义<br>]异常无 | 临床意义<br>□未查<br>临床意义<br>□未查<br>临床意义 |
| 检查项目 红细胞计数(RBC) 白细胞计数(WBC) | | 单位<br>10 <sup>12</sup> /L<br>10 <sup>9</sup> /L | □正常 □ □ □ □ □ □ □ 正常 □ | 意义<br> 异常无<br> 景常无<br> 景常无<br> 景义<br> 异常无 | 临床意义 □未查 临床意义 □未查 临床意义 □未查 临床意义 □未查 |
| 检查项目 红细胞计数(RBC) 白细胞计数(WBC) 血红蛋白(Hb) | | 单位<br>10 <sup>12</sup> /L<br>10 <sup>9</sup> /L<br>g/L<br>10 <sup>9</sup> /L | □正常 □ | 意义<br>章义<br>章 | 临床意义 □未查 临床意义 □未查 临床意义 □未查 临床意义 □未查 |
| 检查项目 红细胞计数(RBC) 白细胞计数(WBC) 血红蛋白(Hb) | | 单位<br>10 <sup>12</sup> /L<br>10 <sup>9</sup> /L<br>g/L | □正常 □ | 异常无<br> 京义<br> 异常之<br> 异常之<br> 异常之<br> 异常无 | 临床意义 □未查 临床意义 临床意义 临床意义 临床意义 临床意义 临床意义 |
| 检查项目 红细胞计数(RBC) 白细胞计数(WBC) 血红蛋白(Hb) | | 单位<br>10 <sup>12</sup> /L<br>10 <sup>9</sup> /L<br>g/L<br>10 <sup>9</sup> /L | □正常 □ □ □ □ □ □ □ 正常 □ | 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 京 </td <td>临床意义</td> <td></td> | 临床意义 |

| 进口细胞汁粉 (I·····) | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
|---------------------------|--------|--------------------|---------------|
| 淋巴细胞计数(Lym) | | 10 /L | □异常有临床意义 □未查 |
| 是否进行血生化检查: □ | 是□否 | | |
| 检查日期: | - - _ | (yyyy-r | nm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| | | □U/L | □正常 □异常无临床意义 |
| 谷丙转氨酶(ALT) | | □IU/L | □异常有临床意义 □未查 |
| 公古北与 h (ACT) | | U/L | □正常 □异常无临床意义 |
| 谷草转氨酶(AST) | | □IU/L | □异常有临床意义 □未查 |
| 石土水井 石米 部会 邢行 (AID) | | U/L | □正常 □异常无临床意义 |
| 碱性磷酸酶(ALP) | | □IU/L | □异常有临床意义 □未查 |
| <b>- A HD /rr 丰 (CTD)</b> | | □umo1/L | □正常 □异常无临床意义 |
| 总胆红素(STB) | | □mg/dl | □异常有临床意义 □未查 |
| 古位阳红丰(DDII) | | umo1/L | □正常 □异常无临床意义 |
| 直接胆红素(DBIL) | | □mg/d1 | □异常有临床意义 □未查 |
| 总蛋白(TP) | | g/L | □正常 □异常无临床意义 |
| 75.25 (17) | | 6/ 2 | □异常有临床意义 □未查 |
| 白蛋白(ALB) g | g/L | □正常 □异常无临床意义 | |
| 727 | | g/ L | □异常有临床意义 □未查 |
| 尿素氮(BUN) | | mmo1/L | □正常 □异常无临床意义 |
| /大乐·· (DOII) | | mmO1/ L | □异常有临床意义 □未查 |
| 血肌酐 (Cr) | | □mg/d1 | □正常 □异常无临床意义 |
| (急性肾衰□是 □否) | | □umo1/L | □异常有临床意义 □未查 |
| 血糖 (Glu) | | mmo1/L | □正常 □异常无临床意义 |
| IIII.17指 (GIU) | | | □异常有临床意义 □未查 |
| 日本(114) | | μ mo1/L | □正常 □异常无临床意义 |
| 尿酸(UA) | | | □异常有临床意义 □未查 |

| £□ (v) | mmo1/L | | □正常 □异常无临床意义 |
|---|---|---|---|
| 钾(K) | | IIIIIO1/L | □异常有临床意义 □未查 |
| 钠(Na) | | mmo1/L | □正常 □异常无临床意义 |
| trj (Na) | | IIIIIO1/L | □异常有临床意义 □未查 |
| 氯(C1) | | mmo1/L | □正常 □异常无临床意义 |
| 录(U1) | | IIIIIO1/L | □异常有临床意义 □未查 |
| 是否进行凝血功能检查: | □是 □否 | | |
| 检查日期: _ | - - _ | (yyyy- <sub>1</sub> | mm-dd) |
| 检查项目 | 检查结果 | 単位 | 临床意义 |
| 海南縣區叶南(DT) | | _ | □正常 □异常无临床意义 |
| 凝血酶原时间(PT) | | S | □异常有临床意义 □未查 |
| 活化部分凝血活酶时间 | | | □正常 □异常无临床意义 |
| (APTT) | | S | □异常有临床意义 □未查 |
| <b>好烧死</b> 点医(p.) | | □g/L | □正常 □异常无临床意义 |
| 纤维蛋白原(Fg) | | □mg/d1 | □异常有临床意义 □未查 |
| 凝血酶时间(TT) | | | □正常 □异常无临床意义 |
| /火 | | S | □异常有临床意义 □未查 |
| D-二聚体(D-Dimer) | | u a /I | □正常 □异常无临床意义 |
| D | 聚体(D-Dimer) μg/L | | □异常有临床意义 □未查 |
| 是否进行血气分析检测: | □是 □否 | | |
| 检查日期: _ | - - _ | (уууу- | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| рН | | | □正常 □异常无临床意义 |
| PI | | | □异常有临床意义 □未查 |
| 血氧饱和度 | | % | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| | | | □正常 □异常无临床意义 |
| 二氧化碳分压(PaCO <sub>2</sub> ) | | mmHg | □异常有临床意义 □未查 |
| 氧分压(PaO <sub>2</sub> ) | | mmHg | □正常 □异常无临床意义 |
| 手(力 /立 (1 aU <sub>2</sub> ) | | iiiiii1g | □异常有临床意义 □未查 |

| 碳酸氢(HCO₃¯) | | mg/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
|---|---|---|---|
| 氧合指数(PaO <sub>2</sub> /FiO <sub>2</sub> ) | | mmHg | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 是否进行血脂检测:□是 | □否 | | |
| 检查日期: | - - | (уууу- | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 总胆固醇(TC) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 甘油三酯(TG) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 高密度脂蛋白(HDL-C) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 低密度脂蛋白(LDL-C) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| | 八、 | 炎症标志 | ————————————————————————————————————— |
| 是否进行炎症标志物检查 | <b>.</b> □是 □否 | | |
| <br> 检查日期: | - - | (уууу- | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| C 反应蛋白 | | □ μ g/L □mg/dl □mg/L | □正常 □异常无临床意义<br>□异常有临床意义 □未查 |
| 降钙素原 | | ng/ml | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| | 九、 | 治疗方象 | ž |
| 新冠感染药物治疗 | | | |
| 来瑞特韦给药情况 | | | |
| 药物规格: _ mg | | | |
| 初始给药日期: _ | _ - | - (y | yyy-mm-dd) |
| 是否持续:□是□□否 | | | |
| 结束给药日期: _ | _ - | - (y | yyy-mm-dd) |
| <br> 给药剂量: _ mg | | | |

| 给药频率: □QD □BID □TID □QW □PRN □其他 |
|------------------------------------------------|
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg |
| 其他新冠治疗药物给药情况 |
| 抗病毒小分子药物 |
| 药物名称:□奈玛特韦片/利托那韦片(Paxlovid)□先诺特韦片/利托那韦片(先诺欣) |
| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德韦片(仁 |
| 明德韦) □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称: □注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径: □□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |

| 中和抗体 |
|-----------------------------------------|
| 药物名称: □COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持:□是 □否 |
| 呼吸支持: □是 □否<br>如"是"请勾选: |

| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
|-------------------------------------------------|
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 十、合并用药 |
| 是否发生合并用药: □是 □否 |
| 如"是"请在此处做药物分类勾选: |
| □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 |
| □抗生素: □抗真菌类 □抗病毒类 |
| □糖皮质激素<br>日期: - (yyyy-mm-dd) |
| 注: 如有合并用药,详细用药请记录在"合并用药记录表" |
| 十一、安全性事件 |
| 是否发生安全性事件: □是 □否 |
| 日期: _ _ - - (yyyy-mm-dd) |
| 注: 如有不良事件,请记录在"不良事件记录表" |
| 十二、疾病诊断信息 |
| 是否确诊新型冠状病毒感染:□是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ - - (yyyy-mm-dd) |
| 入院科室: |

| 是否进入 ICU: □是 □否 |
|----------------------------------|
| 进入日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ - - (yyyy-mm-dd) |
| 是否死亡: □是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |
| 十三、新冠病毒基因检测 |
| 是否保留受试者新冠病毒核酸检测样本:□是□□否 |
| 标本类型:□鼻拭子□咽拭子 |

#### 访视 12-随访期 (第 14 天士2 天)

访视日期: |\_\_|\_|-|\_\_|-|\_| (yyyy-mm-dd) 一、新冠病毒核酸检测\* 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_|\_|-|\_\_|-|\_\_| (yyyy-mm-dd) 标本类型:□鼻咽拭子 □□咽拭子 采样日期: | | | | |-| | | (yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、血氧饱和度 是否进行血氧饱和度检查:□是□□否 检查日期: |\_\_|\_\_|\_\_|-|\_\_|-|\_\_|-|\_\_(yyyy-mm-dd) 单位 检查项目 检查结果 临床意义 □异常无临床意义 □正常 指端脉氧饱和度 □异常有临床意义 □未查 三、生命体征 是否进行生命体征检查:□是□□否 检查日期: | | | | |-| | |-| | (yyyy-mm-dd) 检查项目 检查结果 单位 临床意义 □正常 □异常无临床意义 体温  $^{\circ}$ C □异常有临床意义 □未查 □正常 □异常无临床意义 脉搏 次/分 □异常有临床意义 □未查 □正常 □异常无临床意义 呼吸频率 次/分 □异常有临床意义 □未查

| 血压(收缩压) | | mmHg | □正常 | □异常无临 | 床意义 |
|---|---|---|---|---|---|
| mile (IV-III/II) | | | □异常有□ | 临床意义 | □未查 |
| 血压 (舒张压) | | mmHg | | □异常无临 | |
| | | | □异常有□ | 临床意义 | □未査 |
| | 四、 | 临床症状 | 7 | | |
| 是否有新冠感染相关临床 | 症状:□是 □ | □否 | | | |
| (如"是"),临床症状:[ | □鼻塞或流涕 [ | □咽痛 □ | ]呼吸短促耳 | 或呼吸困难 | □咳嗽 □ |
| 乏力 □肌肉或身体痛 | □头痛 □ | 寒战 □ | 〕发热 □ | ]恶心 □呕鸣 | 止 □腹泻 |
| □嗅觉减退 □味觉减过 | 艮 □其他症状 | : | | | |
| 开始日期: _ _ | - - | _ (yyyy- <u>r</u> | nm-dd) | | |
| 结束日期: _ | - - | _ (yyyy-r | nm-dd) | | |
| | 五、 | 体格检查 | <u> </u> | | |
| 是否进行体格检查:□是 | □否 | | | | |
| 检查日期: _ _ | - - | _ (yyyy-r | nm-dd) | | |
| 检查项目 | 临 | 床意义 | | 若有异常, | ,请描述 |
| 一般情况 | □正常 □∮ | 异常无临床: | 意义 | | |
| /2/113/24 | □异常有临床意 | 义 口: | 未查 | | |
| | □正常 □∮ | 异常无临床 | 意义 | | |
| 2.7 | □异常有临床意 | 义 口: | 未查 | | |
| 胸部 | □正常 □∮ | 异常无临床 | 意义 | | |
| ∀励 日り | | | | | |
| | □异常有临床意 | 义 口: | | | |
| FG か7 | □异常有临床意<br>□正常 □ □ | | 未查 | | |
| 腹部 | | 异常无临床: | 未查<br>意义 | | |
| | □正常 □∮ | 异常无临床: | 未查<br>意义<br>未查 | | |
| 腹部 | □正常 □昇常有临床意 | 异常无临床<br>:义 □<br>异常无临床 | 未查<br>意义<br>未查<br>意义 | | |
| 脊柱和四肢关节 | □正常 □昇常有临床意 | 异常无临床<br>: 义 □ | 未查<br>意义<br>未查<br>意义<br>未查 | | |
| | □正常 □ 5<br>□异常有临床意<br>□正常 □ 5<br>□异常有临床意 | 异常无临床<br>:义 □<br>异常无临床<br>:义 □<br>异常无临床 | 未查<br>意<br>之<br>未查<br>意<br>之<br>未查<br>之<br>未查 | | |
| 脊柱和四肢关节 | □正常 □ | 异常无临床<br>: 义 □ □<br>: 异常无临床<br>: 义 □ □<br>: 异常无临床 | 未 意 来 意 未 意 未 意 未 | | |

| 3 <del>11</del> III | □正常 □ | ]异常无临床 | 意义 |
|---|---|---|---|
| 淋巴 | □异常有临床 | 意义 口 | 未查 |
| 井仙 | □正常 □异常无临床意义 | | |
| | | 意义 口 | 未查 |
| | 六、: | 实验室检 | <u>香</u> # |
| 是否进行血常规检查:□ | 是□否 | | |
| 检查日期: | - - | (yyyy-r | nm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 红细胞计数(RBC) | | $10^{12}/L$ | □正常 □异常无临床意义 |
| 红细胞们致(NDC) | | 10°-/L | □异常有临床意义 □未查 |
| 白细胞计数(WBC) | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
| 口细胞们数(WDC) | | 10°/L | □异常有临床意义 □未查 |
| 血红蛋白(Hb) | | g/L | □正常 □异常无临床意义 |
| 皿红虫口(1110) | | | □异常有临床意义 □未查 |
| 血小板计数(PLT) | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
| 血过气放射 剱(111) | | 10 /L | □异常有临床意义 □未查 |
| 中性粒细胞计数 | | 10 <sup>9</sup> /L | □正常 □异常无临床意义 |
| 门门工作业与山顶区门 致 | | | □异常有临床意义 □未查 |
| 红细胞压积(HCT) | | % | |
| 淋巴细胞计数(Lym) | | 1.00/7 | □正常 □异常无临床意义 |
| 7作□5四旭Ⅵ 致 (LyⅢ) | | 10 <sup>9</sup> /L | □异常有临床意义 □未查 |
| 是否进行血生化检查:□ | 是□否 | | |
| 检查日期: _ _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 谷丙转氨酶(ALT) | | □U/L | □正常 □异常无临床意义 |
| Tryty女(阿(ALI) | | □IU/L | □异常有临床意义 □未查 |
| 谷草转氨酶(AST) | | □U/L | □正常 □异常无临床意义 |

| | □IU/L | □异常有临床意义 □未查 |
|---------------------|-------------------|---------------|
| red to rate was the | □U/L | □正常 □异常无临床意义 |
| 碱性磷酸酶(ALP) | □IU/L | □异常有临床意义 □未查 |
| <b>当田ケま (CTD)</b> | □umo1/L | □正常 □异常无临床意义 |
| 总胆红素 (STB) | □mg/d1 | □异常有临床意义 □未查 |
| 古校明尔丰(DDII) | umo1/L | □正常 □异常无临床意义 |
| 直接胆红素(DBIL) | | □异常有临床意义 □未查 |
| 总蛋白(TP) | g/L | □正常 □异常无临床意义 |
| 心虽日(川) | g/ L | □异常有临床意义 □未查 |
| 白蛋白(ALB) | g/L | □正常 □异常无临床意义 |
| 口蛋口(心的) | g/ L | □异常有临床意义 □未查 |
| 尿素氮 (BUN) | mmo1/L | □正常 □异常无临床意义 |
| /A 系炎( \DUN) | IIIIIO1/L | □异常有临床意义 □未查 |
| 血肌酐 (Cr) | □mg/d1 | □正常 □异常无临床意义 |
| (急性肾衰□是 □否) | □umo1/L | □异常有临床意义 □未查 |
| 血糖(Glu) | mmo1/L | □正常 □异常无临床意义 |
| | | □异常有临床意义 □未查 |
| 尿酸(UA) | μ mol/L | □正常 □异常无临床意义 |
| | μ mo1/ L | □异常有临床意义 □未查 |
| を田 (V) | mmo1/L | □正常 □异常无临床意义 |
| 钾 (K) | IIIIIO1/L | □异常有临床意义 □未查 |
| 钠(Na) | mm o 1 /I | □正常 □异常无临床意义 |
| tyj (Na) | mmo1/L | □异常有临床意义 □未查 |
| 复(01) | mmo1/L | □正常 □异常无临床意义 |
| 氯(C1) | | □异常有临床意义 □未查 |
| 是否进行凝血功能检查:□是 □否 | 是否进行凝血功能检查: □是 □否 | |
| 检查日期: _ _ - - _ | _ (yyyy- | mm-dd) |

| 检查项目 | 检查结果 | 单位 | 临床意义 |
|---|---|---|---|
| | | S | □正常 □异常无临床意义 |
| 凝血酶原时间(PT) | | | □异常有临床意义 □未查 |
| 活化部分凝血活酶时间 | | | □正常 □异常无临床意义 |
| (APTT) | | S | □异常有临床意义 □未查 |
| <b>江州西山田(中)</b> | | g/L | □正常 □异常无临床意义 |
| 纤维蛋白原(Fg) | | □mg/d1 | □异常有临床意义 □未查 |
| | | | □正常 □异常无临床意义 |
| 凝血酶时间(TT) | | S | □异常有临床意义 □未查 |
| D-二聚体(D-Dimer) | | U ~ /I | □正常 □异常无临床意义 |
| D 家体(D-D1mer) | | μg/L | □异常有临床意义 □未查 |
| 是否进行动脉血气分析检 | 测:□是□ | ]否 | |
| 检查日期: _ | - - | (yyyy-r | nm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| | | | □正常 □异常无临床意义 |
| рН | | | □异常有临床意义 □未查 |
| 4. 层 6. 红 6. | | %mmHg | □正常 □异常无临床意义 |
| 血氧饱和度 | | /oiiiiii1g | □异常有临床意义 □未查 |
| 二氧化碳分压 | | mmHg | □正常 □异常无临床意义 |
| 100000 | | o o | □异常有临床意义 □未査 |
| 氧分压 | | mmHg | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 碳酸氢 | | mg/L | □正常 □异常无临床意义 |
| | | | □异常有临床意义 □未查<br>□正常 □异常无临床意义 |
| 氧合指数 | | mmHg | □异常有临床意义 □未查 |
| 是否进行血脂检测: □是 □否 | | | |
| 检查日期: _ _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 总胆固醇(TC) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
| 甘油三酯(TG) | | mmo1/L | □正常 □异常无临床意义 □未查 |

| 高密度脂蛋白(HDL-C) | | mmo1/L | □正常 □异常无临床意义 □异常有临床意义 □未查 |
|---|---|---|---|
| 低密度脂蛋白(LDL-C) | | mmo1/L | □正常 □异常无临床意义 □未查 |
| <br> 是否进行炎症标志物检查 | | <u> </u> | |
| 检查日期: _ | - _ - | (уууу- <sub> </sub> | mm-dd) |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| | | □ µ g/L | |
| C 反应蛋白 | | □mg/d1 | □正常 □异常无临床意义 |
| | | □mg/L | - □异常有临床意义 □未查<br>- □ |
| | | , - | □正常 □异常无临床意义 |
| 降钙素原 | | ng/ml | □异常有临床意义 □未查 |
| | 八、 | 治疗方象 | ₹ |
| 新冠感染药物治疗 | | | |
| 来瑞特韦给药情况 | 来瑞特韦给药情况 | | |
| <br> 药物规格: mg | | | |
| 初始给药日期: _ _ - - (yyyy-mm-dd) | | | |
| 是否持续:□是 □否 | | | |
| 结束给药日期: _ | _ _ - - | - (y | yyy-mm-dd) |
| 给药剂量: _ mg | | | |
| 给药频率:□QD□BID | | QW □PRN | □其他 |
| │<br>│给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | | | |
| <br> 注射 □其他 | | | |
| <br> 总剂量: mg | | | |
| <br> 其他新冠治疗药物给药情 | 其他新冠治疗药物给药情况 | | |
| 抗病毒小分子药物 | | | |
| 药物名称: □奈玛特韦片/利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) | | | |
| <br> □草诺拉韦胶囊(Molnup | iravir) 口阿语 | 兹夫定片 ( 擅 | ▶ (任安) □氢溴酸氘瑞米德韦片(仁 |

| 明德韦) □其他 |
|-----------------------------------------|
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 免疫用药 |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中和抗体 |
| 药物名称:□COVID-19 人免疫球蛋白 □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |

| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
|-------------------------------------------------|
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - _ - _ (yyyy-mm-dd) |
| 是否持续:□是 □否 |
| 结束给药日期: _ - - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗:□是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(FiO2): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |
| 1 |

### 九、合并用药

| 是否发生合并用药:□是 □否 如 "是"请在此处做药物分类勾选:□血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素□抗生素:□抗真菌类 □抗病毒类□糖皮质激素 □期:□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ |
|---|
| 十、安全性事件 |
| 是否发生安全性事件:□是 □否 |
| 日期: _ _ - - (yyyy-mm-dd) |
| 注:如有不良事件,请记录在"不良事件记录表" |
| 十一、疾病诊断信息 |
| 是否确诊新型冠状病毒感染:□是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ _ - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ _ - - (yyyy-mm-dd) |
| 是否入院:□是 □否 |
| 入院日期: _ _ - - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ _ - - (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) |
| 死亡原因: |

#### 访视 13-随访期 (第 28 天士4 天)

访视日期: |\_\_|\_|-|\_\_|-|\_| (yyyy-mm-dd) 一、新冠病毒核酸检测\* 是否进行新冠病毒核酸检测:□是□□否 检测日期: |\_\_|\_|\_|-|\_\_|-|\_|-|(yyyy-mm-dd) 标本类型:□鼻咽拭子 □□咽拭子 采样日期: | | | | |-| | | (yyyy-mm-dd) 新型冠状病毒 ORF1ab 基因: □阴性 □阳性 新型冠状病毒 ORF1ab 基因 Ct 值: 新型冠状病毒 N 基因: □阴性 □阳性 新型冠状病毒 N 基因 Ct 值: 二、胸部影像学检测\* 是否进行胸部影像检查:□是□□否 检查日期: | | | |\_|-|\_|-|\_|-|(yyyy-mm-dd) 检查名称 检查内容 临床意义 □异常无临床意义 □正常 胸部 (肺部) CT □异常有临床意义 □未查 □正常 □异常无临床意义 胸部 (肺部) X 射线 □异常有临床意义 □未查 三、血氧饱和度 是否进行血氧饱和度检查:□是 □否 检查日期: |\_\_|\_|\_|-|\_\_|-|\_|-|\_| (yyyy-mm-dd) 检查项目 检查结果 单位 临床意义 □正常 □异常无临床意义 指端脉氧饱和度 % □异常有临床意义 □未查

| 四、生命体征 | | | |
|---|---|---|---|
| 检查日期: _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 检查结果 | 单位 | 临床意义 |
| 体温 | | °C | □正常 □异常无临床意义 |
| 14-4IIII | | C | □异常有临床意义 □未查 |
| <br> 脉搏 | | 次/分 | □正常 □异常无临床意义 |
| ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | J 4 7 7 | □异常有临床意义 □未查 |
| <br> 呼吸频率 | | 次/分 | □正常 □异常无临床意义 |
| | | · | □异常有临床意义 □未查 |
| 血压(收缩压) | | mmHg | □正常 □异常无临床意义 |
| | | _ | □异常有临床意义 □未查 |
| 血压 (舒张压) | | mmHg | □正常 □异常无临床意义 |
| □异常有临床意义 □未查 | | | |
| 五、临床症状 | | | |
| 是否有新冠感染相关临床 | 症状:□是 □ | □否 | |
| (如"是"),临床症状:□鼻塞或流涕 □咽痛 □呼吸短促或呼吸困难 □咳嗽 □ | | | |
| 乏力 □肌肉或身体痛 □头痛 □寒战 □发热 □恶心 □呕吐 □腹泻 | | | |
| □嗅觉减退 □味觉减退 □其他症状: | | | |
| 开始日期: _ _ | - _ _ | _ (yyyy- <sub>I</sub> | mm-dd) |
| <br> 结束日期: _ _ - - (yyyy-mm-dd) | | | |
| 六、体格检查 | | | |
| 是否进行体格检查:□是 | □否 | | |
| <br> 检查日期: _ - - (yyyy-mm-dd) | | | |
| 检查项目 | 临 | 床意义 | 若有异常,请描述 |
| 一般情况 | □正常□! | 异常无临床 | 意义 |
| AX IH UL | □异常有临床意 | :义 □ | 未查 |
| <br> | □正常 □! | 异常无临床 | 意义 |
| 2 5 7 5 | □异常有临床意 | · Ÿ □ | 未杏 |

| 150 分7 | □正常 □异常无临床意义 |
|---|---|
| 胸部 | □异常有临床意义 □未查 |
| Ff | □正常 □异常无临床意义 |
| 腹部 | □异常有临床意义 □未查 |
| <b>炎</b> 比和Ⅲ肚子芸 | □正常 □异常无临床意义 |
| 脊柱和四肢关节<br> | □异常有临床意义 □未查 |
| 神经系统 | □正常 □异常无临床意义 |
| 押红尔切 | □异常有临床意义 □未查 |
| 皮肤 | □正常 □异常无临床意义 |
| /文/A/X | □异常有临床意义 □未查 |
| 淋巴 | □正常 □异常无临床意义 |
| 717 L | □异常有临床意义 □未查 |
| # 44 | □正常 □异常无临床意义 |
| 其他 | □异常有临床意义 □未查 |
| | 七、治疗方案 |
| 新冠感染药物治疗 | |
| 来瑞特韦给药情况 | |
| 药物规格: mg | |
| 初始给药日期: _ | _ - - (yyyy-mm-dd) |
| 是否持续:□是 □否 | |
| 结束给药日期: _ | _ - - (yyyy-mm-dd) |
| 给药剂量: mg | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 | |
| 注射 □其他 | |
| 总剂量: mg | |
| 其他新冠治疗药物给药情 | 况 |
| 抗病毒小分子药物 | |
| 药物名称:□奈玛特韦片 | /利托那韦片(Paxlovid) □先诺特韦片/利托那韦片(先诺欣) |

| □莫诺拉韦胶囊(Molnupiravir) □阿兹夫定片(捷倍安) □氢溴酸氘瑞米德 | 息韦片 (仁 |
|--------------------------------------------|--------|
| 明德韦) □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ _ - - _ - (yyyy-mm-dd) | |
| 是否持续:□是 □否 | |
| 结束给药日期: _ _ - - _ - (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率: □QD □BID □TID □QW □PRN □其他 | |
| 台药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □胞 | 复膜内药物 |
| 注射 □其他 | |
| 总剂量: mg 或 g | |
| 免疫用药 | |
| 药物名称:□注射用胸腺法新 □糖皮质激素 □白细胞介素 6 抑制剂 □其 | 他 |
| 药物规格: mg 或 g | |
| 初始给药日期: _ _ - - (yyyy-mm-dd) | |
| 是否持续:□是 □否 | |
| 结束给药日期: _ _ - - - (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |
| 给药频率:□QD □BID □TID □QW □PRN □其他 | |
| 恰约途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □№ | 复膜内药物 |
| 注射 □其他 | |
| 总剂量: mg 或 g | |
| 中和抗体 | |
| 药物名称: □COVID-19 人免疫球蛋白 □其他 | |
| 药物规格: mg 或 g | |
| 初始给药日期: _ - - (yyyy-mm-dd) | |
| 是否持续:□是 □否 | |
| 结束给药日期: - - - (yyyy-mm-dd) | |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d | |

| 给药频率: □QD □BID □TID □QW □PRN □其他 |
|-------------------------------------------------|
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 中(成)药 |
| 药物名称:□连花清瘟胶囊 □连花清瘟颗粒 □疏风解毒胶囊 □化湿败毒颗粒 |
| □其他 |
| 药物规格: mg 或 g |
| 初始给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否持续: □是 □否 |
| 结束给药日期: _ - _ - _ - (yyyy-mm-dd) |
| 给药剂量: mg/d 或 g/d 或 mg/kg/d 或 g/kg/d |
| 给药频率: □QD □BID □TID □QW □PRN □其他 |
| 给药途径:□□服 □局部 □舌下给药 □肌肉注射 □静脉输液 □腹膜内药物 |
| 注射 □其他 |
| 总剂量: mg 或 g |
| 新冠非药物干预: |
| 抗凝治疗: □是 □否 |
| 如"是"请勾选:□低分子肝素 □普通肝素 □其他 |
| 呼吸支持: □是 □否 |
| 如"是"请勾选: |
| □鼻导管或面罩吸氧氧疗: |
| 鼻导管吸氧: L/min; 面罩吸氧: L/min; 吸氧浓度(Fi02): %; 小时/天; |
| □高流量湿化氧疗仪经鼻高流量氧疗或无创通气: |
| L/min; ℃; 吸氧浓度 (Fi02): %; 小时/天; |
| 机械通气: □是 □否 |
| 如"是"请勾选:□有创机械通气□体外膜肺氧合无创; |
| 通气模式: ; 潮气量(Vt): ml; 呼吸频率(RR): 次/分; |
| 呼气末正压 (PEEP): cmH20; 吸氧浓度 (Fi02): %; 小时/天; |

| 八、合并用药 |
|---|
| 是否发生合并用药:□是 □否 如"是"请在此处做药物分类勾选: □血管活性药物:□多巴胺 □肾上腺素 □去甲肾上腺素 □抗生素:□抗真菌类 □抗病毒类 □糖皮质激素 日期: (yyyy-mm-dd) 注:如有合并用药,详细用药请记录在"合并用药记录表" |
| 九、安全性事件 |
| 是否发生安全性事件:□是 □否 □用: _ _ - - (yyyy-mm-dd) 注: 如有不良事件,请记录在"不良事件记录表" |
| 十、疾病诊断信息 |
| 是否确诊新型冠状病毒感染:□是 □否 |
| 确诊方式:□流行病学史 □临床表现 □核酸检测 □其他 |
| 确诊日期: _ - - - (yyyy-mm-dd) |
| 新型冠状病毒感染分型:□轻型 □中型 □重型 □危重型 |
| 是否确诊脓毒症:□是 □否 |
| (如"是"), SOFA 评分: |
| 确诊日期: _ - - - (yyyy-mm-dd) |
| 是否入院: □是 □否 |
| 入院日期: _ - _ - _ - (yyyy-mm-dd) |
| 入院科室: |
| 是否进入 ICU: □是 □否 |
| 进入日期: _ _ - - (yyyy-mm-dd) |
| 是否出院:□是 □否 |
| 出院日期: _ - _ - _ - (yyyy-mm-dd) |
| 是否死亡:□是 □否 |
| 死亡日期: _ _ - - (yyyy-mm-dd) 死亡原因: |

# 计划外访视

| 访视日期: - - - - - - - (yyyy-mm- |
|-----------------------------------|
|-----------------------------------|

| 检查项目 | 检查日期<br>(yyyy-mm-dd) | 结果描述<br>(实验室检查需注明单位) | 临床意义 | 检查目的 |
|------|----------------------|----------------------|----------------|------|
| | | | □正常 | |
| | | | <br> □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常, 无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |
| | | | □正常 | |
| | | | □异常,无临床意义 | |
| | | | □异常,有临床意义 | |

## 合并用药记录表

#### 在试验期间是否有合并用药: □是 □否, (如"是"),请填写在下表:

| 药物名称 | 药物 分类 | 给药 途径 | 每次剂量<br>(注明单<br>位) | 给药频率 | 开始日期<br>(yyyy-mm-dd) | 是否持续 | 结束日期<br>(yyyy-mm-d<br>d) | 用药原因 |
|---|---|---|---|---|---|---|---|---|
| | | | | | | □是□否 | | |

## 不良反应(AE)记录表

#### 受试者姓名拼音缩写: |\_\_|\_\_|\_\_|

| AE<br>名称 | 分级<br>(CTCAE 分级) | PARTICIPATION TO THE PARTICIPATION OF THE PARTICIPA | 分级 开始日期 结束日期 与研究药物关系 | 是否导致 是否有 | 对试验用药采取措施 | *+.17 | 签名 | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | (yyyy-mm-dd) | 来瑞特韦片 | SAE | 纠正治疗 | 来瑞特韦片 | 转归 | 金色 |
| | □I級 □II級<br>□III级 □IV级<br>□V级 | | | 口肯定有关 口可能有关<br>口可能无关 口肯定无关<br>口无法判定 | □是□否 | □是□□否 | 口暂缓给药 口停止给药<br>口终止试验 口不适用<br>口未知 | □未恢复/未解决 □恢复/解决 □恢复/解决后有后遗症 □缓解 □加重 □死亡 □未知 | |
| | □I級 □II級<br>□III級 □IV級<br>□V級 | | | 口肯定有关 口可能有关<br>口可能无关 口肯定无关<br>口无法判定 | 口是口否 | □是□否 | 口暂缓给药 口停止给药<br>口终止试验 口不适用<br>口未知 | □未恢复/未解决 □恢复/解决 □恢复/解决后有后遗症 □缓解 □加重 □死亡 □未知 | |
| | □I级 □II级<br>□III级 □IV级<br>□V级 | | | 口肯定有关 口可能有关<br>口可能无关 口肯定无关<br>口无法判定 | 口是口否 | 口是口否 | 口暂缓给药 口停止给药<br>口终止试验 口不适用<br>口未知 | □未恢复/未解决 □恢复/解决 □恢复/解决后有后遗症 □缓解 □加重 □死亡 □未知 | |
| | □I級 □II級<br>□III級 □IV級<br>□V級 | | | 口肯定有关 口可能有关<br>口可能无关 口肯定无关<br>口无法判定 | 口是口否 | 口是口否 | 口暂缓给药 口停止给药<br>口终止试验 口不适用<br>口未知 | □未恢复/未解决 □恢复/解决 □恢复/解决后有后遗症 □缓解 □加重 □死亡 □未知 | |

### 严重不良事件报告表(SAE)

## 受试者姓名拼音缩写: |\_\_|\_\_|\_\_|

| 报告类型 | □首次报告 □随访报告 □总结报告 |
|---|---|
| 首次报告日期: _ | - - (yyyy-mm-dd) |
| 总结报告日期: _ | _ _ - _ - _ (yyyy-mm-dd) |
| SAE 名称 | |
| SAE 情况 | □导致住院 □延长住院时间 □伤残 □功能障碍 □导致先天畸形 □危及生命或死亡 □其它: |
| SAE 发生时间: _ | _ - - (yyyy-mm-dd) |
| SAE 反应严重程度 | □轻度 □中度 □重度 |
| 对试验用药采取的措施 | □剂量不变 □暂停给药 □暂停给药后又恢复 |
| <b>刈风</b> 湿用约木取的相胞 | □剂量下调 □终止给药 |
| SAE 转归 | □症状消失(后遗症□有 □无) □症状持续 |
| <b>2.5</b> 上 上 水 大 大 女 头 ズ | □死亡 (死亡时间: _ _ - _ - _ - _ (yyyy-mm-dd)) |
| SAE 与试验药的关系 | □肯定有关 □很可能有关 □可能有关 □可能无关 □肯定无关 |
| SAE 报道情况 | 国内: □有 □无 □不详 |
| 0.15 1K/C 100 | 国外:□有 □无 □不详 |
| SAE 发生及处理的详细情 | 况(首次报告): |
| SAE 发生及处理的详细情 | 况(随访报告 1): |
| SAE 发生及处理的详细情况(随访报告 2): | |
| SAE 发生及处理的详细情 | 况(总结报告): |

# 研究总结

## 受试者姓名拼音缩写: |\_\_|\_\_|\_\_|

| 是否按方案要求完成本项临床试验 | □是 □否 |
|-------------------------|-----------------------------------|
| 如完成试验, | |
| 完成试验日期: _ _ - _ - _ · | - (yyyy-mm-dd) |
| 如未完成试验, | |
| 终止试验日期: _ _ - _ - _ · | - (yyyy-mm-dd) |
| 末次访视日期: _ _ - - | - (yyyy-mm-dd) |
| 试验期间是否有终点事件发生:□是 | □否 |
| 试验期间是否有不良事件发生:□是 | □否 |
| 首先提出中止试验的是:□受试者 □ | 试验研究者 □项目管理部门 □其它: |
| 受试者退出研究的原因: | |
| □发生严重不良事件 □受试者怀孕 | □同时参加其他临床研究 □受试者要求退出 |
| □研究者认为需要中止试验 □其它: | |
| 研究者签名: | 签署日期: _ _ - - _ - (yyyy-mm-dd) |

#### 病例报告表(CRF)审核声明

本试验中心负责人特此声明,经审核,此病例报告中所有项目的记录都是真实、准确的。

| 试验中心负责人 | 、签名: | | |
|---------|------|---|---|
| 日期: | 年 | 月 | 日 |

本人作为该研究监查员特此声明,经审核,此病例报告表中所有项目的记录与原始病历相符,是真实、完整和准确的。